CLINICAL TRIAL: NCT04425629
Title: A Master Protocol Assessing the Safety, Tolerability, and Efficacy of Anti-Spike (S) SARS-CoV-2 Monoclonal Antibodies for the Treatment of Ambulatory Patients With COVID-19
Brief Title: Safety, Tolerability, and Efficacy of Anti-Spike (S) SARS-CoV-2 Monoclonal Antibodies for the Treatment of Ambulatory Adult and Pediatric Patients With COVID-19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Emerging SARS-CoV-2 variants impacting susceptibility to study drug
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R10933-10987-COV-2067; 2020-003690-21 (EudraCT Number)
Expanded Access: NCT04617535 (No longer available)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-COV-2); coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — casirivimab and imdevimab drug combination; casirivimab; imdevimab

STUDY DESIGN:
Intervention Model Description: Phase 1/Phase 2/Phase 3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- casirivimab+imdevimab low dose (Experimental): Low dose or body-weight equivalent for those under 18 years of age.
  Interventions: Drug: casirivimab+imdevimab combination therapy

INTERVENTIONS:
Drug: casirivimab+imdevimab combination therapy — Administered intravenously (IV) single dose
  Other Names: REGN-COV2; REGN10933; REGN10987; REGEN-COV™; Ronapreve™

SUMMARY:
Phase 1

* To evaluate the safety and tolerability of REGN10933+REGN10987 compared to placebo
* To evaluate the virologic efficacy of REGN10933+REGN10987 compared to placebo in reducing viral load of SARS-CoV-2

Phase 2

• To evaluate the virologic efficacy of REGN10933+REGN10987 compared to placebo in reducing viral load of SARS-CoV-2

Phase 3

* Cohort 1 (≥18 Years Old, Not Pregnant at Randomization)

  • To evaluate the clinical efficacy of REGN10933+REGN10987 compared to placebo as measured by COVID-19-related hospitalizations or all-cause death
* Cohort 2 (<18 Years Old, Not Pregnant at Randomization)

  * To evaluate the safety and tolerability of REGN10933+REGN10987 compared to placebo
  * To further characterize the concentrations of REGN10933 and REGN10987 in serum over time
* Cohort 3 (Pregnant at Randomization) • To evaluate the safety and tolerability of REGN10933+REGN10987

ELIGIBILITY:
Key Inclusion Criteria:

* Has SARS-CoV-2-positive diagnostic test (from a sample collected ≤72 hours prior to randomization, using a validated SARS-CoV-2 antigen, RT-PCR, or other molecular diagnostic assay, and an appropriate sample such as nasopharyngeal [NP], nasal, oropharyngeal [OP], or saliva)
* Has symptoms consistent with COVID-19, as determined by the investigator, with onset ≤7 days before randomization
* Maintains O2 saturation ≥93% on room air
* Is able to understand and complete study-related questionnaires (patients aged ≥12 years only)

Key Exclusion Criteria:

* Was admitted to a hospital for COVID-19 prior to randomization, or is hospitalized (inpatient) for any reason at randomization
* Has participated, or is participating, in a clinical research study evaluating COVID-19 convalescent plasma, mAbs against SARS-CoV-2 (eg, bamlanivimab), or intravenous immunoglobulin (IVIG) within 3 months or within 5 half-lives of the investigational product (whichever is longer) prior to the screening visit
* Prior, current, or planned future use of any of the following treatments: COVID-19 convalescent plasma, mAbs against SARS-CoV-2 (eg, bamlanivimab), IVIG (any indication), systemic corticosteroids (any indication), or COVID-19 treatments (authorized, approved, or investigational)
* Prior use (prior to randomization), current use (at randomization) or planned use (within 90 days of study drug administration or per current CDC recommendations, as applicable) of any authorized or approved vaccine for COVID-19
* Has participated, is participating or plans to participate in a clinical research study evaluation any authorized, approved or investigational vaccine for COVID-19

NOTE: Other Protocol defined Inclusion/Exclusion criteria apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10078 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (91):
- United States (81):
  - Regeneron Study Site, Mesa, Arizona
  - Regeneron Study Site, Tucson, Arizona
  - Regeneron Study Site, Canoga Park, California
  - Regeneron Study Site, La Mesa, California
  - Regeneron Study Site, La Palma, California
  - Regeneron Study Site 1, Long Beach, California
  - Regeneron Study Site 2, Long Beach, California
  - Regeneron Study Site 3, Long Beach, California
  - Regeneron Study Site, Los Angeles, California
  - Regeneron Study Site, Montclair, California
  - Regeneron Study Site, Rolling Hills Estates, California
  - Regeneron Study Site, Sacramento, California
  - Regeneron Study Site, San Francisco, California
  - Regeneron Study Site, Santa Monica, California
  - Regeneron Study Site, Stanford, California
  - Regeneron Study Site, Aurora, Colorado
  - Regeneron Study Site, Colorado Springs, Colorado
  - Regeneron Study Site, Washington D.C., District of Columbia
  - Regeneron Study Site, Boca Raton, Florida
  - Regeneron Study Site, DeLand, Florida
  - Regeneron Study Site, Ft. Pierce, Florida
  - Regeneron Study Site, Hialeah, Florida
  - Regeneron Study Site, Loxahatchee Groves, Florida
  - Regeneron Study Site, Maitland, Florida
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site 1, Miami, Florida
  - Regeneron Study Site 2, Miami, Florida
  - Regeneron Study Site, Sarasota, Florida
  - Regeneron Study Site, St. Petersburg, Florida
  - Regeneron Study Site, Tampa, Florida
  - Regeneron Study Site, West Palm Beach, Florida
  - Regeneron Study Site, Winter Haven, Florida
  - Regeneron Study Site, Winter Park, Florida
  - Regeneron Study Site, Atlanta, Georgia
  - Regeneron Study Site, Augusta, Georgia
  - Regeneron Study Site, Columbus, Georgia
  - Regeneron Study Site, Marietta, Georgia
  - Regeneron Study Site, Chicago, Illinois
  - Regeneron Study Site 1, Downers Grove, Illinois
  - Regeneron Study Site 2, Downers Grove, Illinois
  - Regeneron Study Site, Downers Grove, Illinois
  - Regeneron Study Site, Ames, Iowa
  - Regeneron Study Site, Iowa City, Iowa
  - Regeneron Study Site, Lake Charles, Louisiana
  - Regeneron Study Site, Marrero, Louisiana
  - Regeneron Study Site, New Orleans, Louisiana
  - Regeneron Study Site, Shreveport, Louisiana
  - Regeneron Study Site, Baltimore, Maryland
  - Regeneron Study Site, Royal Oak, Michigan
  - Regeneron Study Site, Jackson, Mississippi
  - Regeneron Study Site, Las Vegas, Nevada
  - Regeneron Study Site, Ridgewood, New Jersey
  - Regeneron Study Site, Teaneck, New Jersey
  - Regeneron Study Site, Santa Fe, New Mexico
  - Regeneron Study Site, Jamaica, New York
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, The Bronx, New York
  - Regeneron Study Site, Charlotte, North Carolina
  - Regeneron Study Site, Durham, North Carolina
  - Regeneron Study Site, Wilmington, North Carolina
  - Regeneron Study Site, Columbus, Ohio
  - Regeneron Study Site, Dayton, Ohio
  - Regeneron Study Site, Philadelphia, Pennsylvania
  - Regeneron Study Site, Providence, Rhode Island
  - Regeneron Study Site, Charleston, South Carolina
  - Regeneron Study Site, Clinton, South Carolina
  - Regeneron Study Site, Sioux Falls, South Dakota
  - Regeneron Study Site 2, Memphis, Tennessee
  - Regeneron Study Site, Memphis, Tennessee
  - Regeneron Study Site, Amarillo, Texas
  - Regeneron Study Site, Corpus Christi, Texas
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, Pearland, Texas
  - Regeneron Study Site, Red Oak, Texas
  - Regeneron Study Site, San Antonio, Texas
  - Regeneron Study Site, Tyler, Texas
  - Regeneron Study Site, Falls Church, Virginia
  - Regeneron Study Site, Everett, Washington
  - Regeneron Study Site, Seattle, Washington
  - Regeneron Study Site, Madison, Wisconsin
- Mexico (9):
  - Regeneron Study Site, Guadalajara, Jalisco
  - Regeneron Study Site, Zapopan, Jalisco
  - Regeneron Study Site, Monterrey, Nuevo León
  - Regeneron Study Site, Mérida, Yucatán
  - Regeneron Study Site, Chihuahua City
  - Regeneron Study Site, Durango
  - Regeneron Study Site, Mexico City
  - Regeneron Study Site, Mérida
  - Regeneron Study Site, Veracruz
- Regeneron Study Site, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., Food and Drug Administration (FDA), European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- [Derived] Norton TD, Thakur M, Ganguly S, Ali S, Chao J, Waldron A, Xiao J, Patel Y, Turner KC, Davis JD, Irvin SC, Pan C, Atmodjo-Watkins D, Hooper AT, Hamilton JD, Subramaniam D, Bocchini JA, Kowal B, DiCioccio AT, Bhore R, Geba GP, Cox E, Braunstein N, Dakin P, Herman GA. Assessing the safety and pharmacokinetics of casirivimab and imdevimab (CAS+IMD) in a cohort of pregnant outpatients with COVID-19: results from an adaptive, multicentre, randomised, double-blind, phase 1/2/3 study. BMJ Open. 2024 Oct 8;14(10):e087431. doi: 10.1136/bmjopen-2024-087431. PMID 39384241
- [Derived] Rofail D, Hussein M, Naumann U, Podolanczuk AJ, Norton T, Ali S, Mastey V, Ivanescu C, Hirshberg B, Geba GP. Patient-Reported Outcomes in COVID-19 Treatment with Monoclonal Antibodies Reveal Benefits in Return to Usual Activities. Infect Dis Ther. 2024 Aug;13(8):1861-1876. doi: 10.1007/s40121-024-01013-1. Epub 2024 Jul 3. PMID 38961047
- [Derived] Bermejo-Gomez A, Aguilera-Alonso D, Rincon-Lopez EM, Catalan-Alonso P, Bardon-Cancho EJ, Garcia-Morin M, Manrique-Rodriguez S, Navarro-Gomez ML. Use of Monoclonal Antibodies in a Pediatric Patient With Severe Combined Immunodeficiency and Persistent SARS-CoV-2 Infection. Pediatr Infect Dis J. 2023 Aug 1;42(8):e290-e292. doi: 10.1097/INF.0000000000003938. Epub 2023 Apr 27. PMID 37079569
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Weinreich DM, Sivapalasingam S, Norton T, Ali S, Gao H, Bhore R, Xiao J, Hooper AT, Hamilton JD, Musser BJ, Rofail D, Hussein M, Im J, Atmodjo DY, Perry C, Pan C, Mahmood A, Hosain R, Davis JD, Turner KC, Baum A, Kyratsous CA, Kim Y, Cook A, Kampman W, Roque-Guerrero L, Acloque G, Aazami H, Cannon K, Simon-Campos JA, Bocchini JA, Kowal B, DiCioccio AT, Soo Y, Geba GP, Stahl N, Lipsich L, Braunstein N, Herman G, Yancopoulos GD; Trial Investigators. REGEN-COV Antibody Combination and Outcomes in Outpatients with Covid-19. N Engl J Med. 2021 Dec 2;385(23):e81. doi: 10.1056/NEJMoa2108163. Epub 2021 Sep 29. PMID 34587383
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Weinreich DM, Sivapalasingam S, Norton T, Ali S, Gao H, Bhore R, Musser BJ, Soo Y, Rofail D, Im J, Perry C, Pan C, Hosain R, Mahmood A, Davis JD, Turner KC, Hooper AT, Hamilton JD, Baum A, Kyratsous CA, Kim Y, Cook A, Kampman W, Kohli A, Sachdeva Y, Graber X, Kowal B, DiCioccio T, Stahl N, Lipsich L, Braunstein N, Herman G, Yancopoulos GD; Trial Investigators. REGN-COV2, a Neutralizing Antibody Cocktail, in Outpatients with Covid-19. N Engl J Med. 2021 Jan 21;384(3):238-251. doi: 10.1056/NEJMoa2035002. Epub 2020 Dec 17. PMID 33332778

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10065 were randomized, 135 randomized but not treated
Groups:
- Phase 1 Symptomatic: Placebo; Phase 2 Symptomatic: Placebo: Placebo of R10933 + R10987 Adult Symptomatic Participants with COVID-19
- Phase 1 Symptomatic: 2.4 IV; Phase 2 Symptomatic: 2.4 IV: 2.4g of R10933 + R10987 Adult Symptomatic Participants with COVID-19
- Phase 1 Symptomatic: 8.0 IV; Phase 2 Symptomatic: 8.0 IV: 8.0g of R10933 + R10987 Adult Symptomatic Participants with COVID-19
- Phase 2 Asymptomatic: Placebo: Placebo of R10933 + R10987 Adult Participants with asymptomatic SARS-CoV-2 infection
- Phase 2 Asymptomatic: 2.4 IV: 2.4g of R10933 + R10987 Adult Participants with asymptomatic SARS-CoV-2 infection
- Phase 2 Asymptomatic: 8.0 IV: 8.0g of R10933 + R10987 Adult Participants with asymptomatic SARS-CoV-2 infection
- Phase 3 Age>=18: Placebo: Placebo of R10933 + R10987 Participants >= 18 with COVID-19, not pregnant at randomization
- Phase 3 Age>=18: 1.2 IV: 1.2g of R10933 + R10987 Participants >= 18 with COVID-19, not pregnant at randomization
- Phase 3 Age>=18: 2.4 IV: 2.4g of R10933 + R10987 Participants >= 18 with COVID-19, not pregnant at randomization
- Phase 3 Age>=18: 8.0 IV: 8.0g of R10933 + R10987 Participants >= 18 with COVID-19, not pregnant at randomization
- Phase 3 Age <18: Placebo: Placebo of R10933 + R10987 Participants <18 with COVID-19, not pregnant at randomization
- Phase 3 Age <18: 1.2 IV: 1.2g of R10933 + R10987 Participants <18 with COVID-19
- Phase 3 Age <18: 2.4 IV: 2.4g of R10933 + R10987 Participants <18 with COVID-19
- Phase 3 Pregnant Placebo: Placebo of R10933 + R10987 Participants who are pregnant with COVID-19
- Phase 3 Pregnant 1.2 IV: 1.2g of R10933 + R10987 Participants who are pregnant with COVID-19
- Phase 3 Pregnant: 2.4 IV: 2.4g of R10933 + R10987 Participants who are pregnant with COVID-19
Period: Overall Study
Arm/Group | Phase 1 Symptomatic: Placebo | Phase 1 Symptomatic: 2.4 IV | Phase 1 Symptomatic: 8.0 IV | Phase 2 Symptomatic: Placebo | Phase 2 Symptomatic: 2.4 IV | Phase 2 Symptomatic: 8.0 IV | Phase 2 Asymptomatic: Placebo | Phase 2 Asymptomatic: 2.4 IV | Phase 2 Asymptomatic: 8.0 IV | Phase 3 Age>=18: Placebo | Phase 3 Age>=18: 1.2 IV | Phase 3 Age>=18: 2.4 IV | Phase 3 Age>=18: 8.0 IV | Phase 3 Age <18: Placebo | Phase 3 Age <18: 1.2 IV | Phase 3 Age <18: 2.4 IV | Phase 3 Pregnant Placebo | Phase 3 Pregnant 1.2 IV | Phase 3 Pregnant: 2.4 IV
Started | 24 | 24 | 24 | 242 | 242 | 243 | 76 | 76 | 76 | 2378 | 2156 | 3189 | 1027 | 2 | 129 | 75 | 3 | 43 | 36
Completed | 23 | 19 | 22 | 230 | 232 | 233 | 71 | 73 | 74 | 2217 | 1974 | 2947 | 962 | 2 | 123 | 65 | 2 | 40 | 33
Not Completed | 1 | 5 | 2 | 12 | 10 | 10 | 5 | 3 | 2 | 161 | 182 | 242 | 65 | 0 | 6 | 10 | 1 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 1 | 7 | 1 | 2 | 1 | 0 | 1 | 64 | 70 | 98 | 30 | 0 | 5 | 4 | 0 | 3 | 1
Not completed — Subject Decision | 0 | 2 | 1 | 3 | 6 | 6 | 3 | 3 | 1 | 70 | 95 | 124 | 25 | 0 | 1 | 4 | 1 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Request | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 0 | 0 | 9 | 9 | 10 | 8 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 5 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 3 Age>=18: Placebo: Placebo of R10933 + R10987 Participants >=18 with COVID-19, not pregnant at randomization
- Phase 3 Age>=18: 1.2 IV: 1.2g of R10933 + R10987 Participants >=18 with COVID-19, not pregnant at randomization
- Phase 3 Age>=18: 2.4 IV: 2.4g of R10933 + R10987 Participants >=18 with COVID-19, not pregnant at randomization
- Phase 3 Age>=18: 8.0 IV: 8.0g of R10933 + R10987 Participants >=18 with COVID-19, not pregnant at randomization
- Total: Total of all reporting groups
Arm/Group | Phase 1 Symptomatic: Placebo | Phase 1 Symptomatic: 2.4 IV | Phase 1 Symptomatic: 8.0 IV | Phase 2 Symptomatic: Placebo | Phase 2 Symptomatic: 2.4 IV | Phase 2 Symptomatic: 8.0 IV | Phase 2 Asymptomatic: Placebo | Phase 2 Asymptomatic: 2.4 IV | Phase 2 Asymptomatic: 8.0 IV | Phase 3 Age>=18: Placebo | Phase 3 Age>=18: 1.2 IV | Phase 3 Age>=18: 2.4 IV | Phase 3 Age>=18: 8.0 IV | Phase 3 Age <18: Placebo | Phase 3 Age <18: 1.2 IV | Phase 3 Age <18: 2.4 IV | Phase 3 Pregnant Placebo | Phase 3 Pregnant 1.2 IV | Phase 3 Pregnant: 2.4 IV | Total
Number analyzed (Participants) | 24 | 24 | 24 | 242 | 242 | 243 | 76 | 76 | 76 | 2378 | 2156 | 3189 | 1027 | 2 | 129 | 75 | 3 | 43 | 36 | 10065
Age, Continuous [Median (Full Range); unit: years] | 40.5 [18 to 72] | 39.5 [18 to 65] | 39.0 [20 to 72] | 42.0 [18 to 89] | 43.0 [18 to 85] | 42.0 [19 to 80] | 43.5 [18 to 80] | 44.5 [18 to 75] | 44.5 [18 to 84] | 46.0 [18 to 92] | 48.0 [18 to 93] | 46.0 [18 to 96] | 44.0 [18 to 90] | 14.0 [12 to 16] | 11.0 [0 to 17] | 12.0 [3 to 17] | 33.0 [27 to 33] | 30.0 [19 to 41] | 28.0 [17 to 41] | 45.0 [0 to 96]
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 129 | 75 | 0 | 0 | 1 | 207
  >=18, <65 | 22 | 23 | 23 | 226 | 223 | 228 | 71 | 62 | 65 | 2159 | 1937 | 2843 | 911 | 0 | 0 | 0 | 3 | 43 | 35 | 8874
  >=65 | 2 | 1 | 1 | 16 | 19 | 15 | 5 | 14 | 11 | 219 | 219 | 346 | 116 | 0 | 0 | 0 | 0 | 0 | 0 | 984
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 10 | 122 | 130 | 136 | 40 | 37 | 32 | 1227 | 1117 | 1635 | 518 | 2 | 69 | 22 | 3 | 43 | 36 | 5203
  Male | 14 | 10 | 14 | 120 | 112 | 107 | 36 | 39 | 44 | 1151 | 1039 | 1554 | 509 | 0 | 60 | 53 | 0 | 0 | 0 | 4862
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 30 | 72 | 84 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 197
  Asian | 0 | 0 | 0 | 4 | 6 | 4 | 1 | 4 | 3 | 89 | 71 | 96 | 45 | 0 | 1 | 1 | 0 | 0 | 0 | 325
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 6 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 17
  Black or African American | 3 | 7 | 0 | 21 | 20 | 23 | 6 | 3 | 5 | 110 | 112 | 172 | 46 | 1 | 8 | 7 | 1 | 4 | 2 | 551
  White | 20 | 16 | 23 | 207 | 208 | 207 | 65 | 69 | 65 | 2010 | 1704 | 2612 | 889 | 1 | 115 | 63 | 2 | 35 | 33 | 8344
  More than one race | 0 | 0 | 0 | 3 | 1 | 3 | 2 | 0 | 3 | 82 | 138 | 143 | 21 | 0 | 3 | 2 | 0 | 1 | 0 | 402
  Unknown or Not Reported | 0 | 1 | 1 | 5 | 6 | 5 | 2 | 0 | 0 | 54 | 52 | 76 | 21 | 0 | 2 | 2 | 0 | 1 | 1 | 229
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 17 | 129 | 121 | 117 | 34 | 43 | 35 | 1002 | 1140 | 1413 | 316 | 0 | 87 | 40 | 0 | 6 | 8 | 4527
  Not Hispanic or Latino | 16 | 12 | 6 | 112 | 121 | 126 | 40 | 33 | 39 | 1357 | 992 | 1740 | 701 | 2 | 42 | 33 | 2 | 37 | 28 | 5439
  Not Reported | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 19 | 24 | 36 | 10 | 0 | 0 | 2 | 1 | 0 | 0 | 99
Race [Count of Participants; unit: Participants]
  White | 20 | 16 | 23 | 207 | 208 | 207 | 65 | 69 | 65 | 2010 | 1704 | 2612 | 889 | 1 | 115 | 63 | 2 | 35 | 33 | 8344
  Black or African American | 3 | 7 | 0 | 21 | 20 | 23 | 6 | 3 | 5 | 110 | 112 | 172 | 46 | 1 | 8 | 7 | 1 | 4 | 2 | 551
  Asian | 0 | 0 | 0 | 4 | 6 | 4 | 1 | 4 | 3 | 89 | 71 | 96 | 45 | 0 | 1 | 1 | 0 | 0 | 0 | 325
  American Indian or Alaska Native | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 30 | 72 | 84 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 197
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 6 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 17
  Unknown | 0 | 0 | 0 | 3 | 1 | 3 | 2 | 0 | 3 | 82 | 138 | 143 | 21 | 0 | 3 | 2 | 0 | 1 | 0 | 402
  Not Reported | 0 | 1 | 1 | 5 | 6 | 5 | 2 | 0 | 0 | 54 | 52 | 76 | 21 | 0 | 2 | 2 | 0 | 1 | 1 | 229
Age Continous [Mean (Standard Deviation); unit: years] | 43.8 (14.42) | 38.9 (11.11) | 40.4 (11.83) | 42.5 (15.21) | 42.7 (15.59) | 41.7 (14.38) | 43.5 (15.51) | 44.8 (16.70) | 44.0 (17.43) | 45.4 (14.61) | 46.7 (14.59) | 46.1 (14.89) | 44.8 (15.09) | 14.0 (2.83) | 10.9 (4.14) | 12.2 (3.36) | 31.0 (3.46) | 28.9 (5.87) | 28.3 (6.02) | 44.7 (15.51)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs) - [Ph1, Ph2, Ph3 Cohort 1 - Cohort 3]
Description: Primary:
  Phase 1, Phase 3 (Cohort 2 and Cohort 3)
  Secondary:
  Phase 2, Phase 3 (Cohort 1)
Time Frame: Through Day 29
Population: Analysis populations were prespecified in the SAP. Pooled analyses were performed for symptomatic adult participants randomized in Phase 1, 2, or 3 (cohort 1) on or before 2/24/21 to placebo, R10933+R10987 1.2 g, 2.4 g, or 8.0 g IV. No phase 1 or 2 participants were randomized to R10933+R10987 1.2 g IV. Asymptomatic adult participants randomized to the asymptomatic cohort of phase 2, symptomatic pediatric / pregnant participants randomized in phase 3 to cohort 2 or 3 were analyzed separately
Measure: Count of Participants; unit: Participants
Groups:
- Combined Phases 1, 2, & 3 Cohort 1 Symptomatic (Placebo): Placebo of R10933 + R10987 Adult Symptomatic Participants with COVID-19
- Combined Phases 1, 2, & 3 Cohort 1 Symptomatic (2.4 IV): Pooled analysis of Phases 1, 2, & 3 Cohort 1 Symptomatic Participants for dosage of 2.4g IV
- Combined Phases 1, 2, & 3 Cohort 1 Symptomatic (8.0 IV): Pooled analysis of Phases 1, 2, & 3 Cohort 1 Symptomatic Participants for dosage of 8.0g IV
- Phase 2 Asymptomatic (Placebo): Placebo of R10933 + R10987 Adult Participants with asymptomatic SARS-CoV-2 infection
- Phase 2 Asymptomatic (2.4g IV): 2.4g of R10933 + R10987 Adult Participants with asymptomatic SARS-CoV-2 infection
- Phase 2 Asymptomatic (8.0g IV): 8.0g of R10933 + R10987 Adult Participants with asymptomatic SARS-CoV-2 infection
- Phase 3 Cohort 1 (1.2g IV) Symptomatic: Phase 3 Cohort 1(1.2g IV) Symptomatic Participants
- Phase 3 Cohort 2 Pediatric (Placebo): Phase 3 Cohort 2 Pediatric (Placebo)
- Phase 3 Cohort 2 Pediatric (1.2g IV): Phase 3 Cohort 2 Pediatric (1.2g IV)
- Phase 3 Cohort 2 Pediatric (2.4g IV): Phase 3 Cohort 2 Pediatric (2.4g IV)
- Phase 3 Cohort 3 Pregnant (Placebo): Phase 3 Cohort 3 Pregnant (Placebo)
- Phase 3 Cohort 3 Pregnant (1.2g IV): Phase 3 Cohort 3 Pregnant (1.2g IV)
- Phase 3 Cohort 3 Pregnant (2.4g IV): Phase 3 Cohort 3 Pregnant (2.4g IV)
Arm/Group | Combined Phases 1, 2, & 3 Cohort 1 Symptomatic (Placebo) | Combined Phases 1, 2, & 3 Cohort 1 Symptomatic (2.4 IV) | Combined Phases 1, 2, & 3 Cohort 1 Symptomatic (8.0 IV) | Phase 2 Asymptomatic (Placebo) | Phase 2 Asymptomatic (2.4g IV) | Phase 2 Asymptomatic (8.0g IV) | Phase 3 Cohort 1 (1.2g IV) Symptomatic | Phase 3 Cohort 2 Pediatric (Placebo) | Phase 3 Cohort 2 Pediatric (1.2g IV) | Phase 3 Cohort 2 Pediatric (2.4g IV) | Phase 3 Cohort 3 Pregnant (Placebo) | Phase 3 Cohort 3 Pregnant (1.2g IV) | Phase 3 Cohort 3 Pregnant (2.4g IV)
Number analyzed (Participants) | 2609 | 2614 | 1272 | 74 | 72 | 73 | 1329 | 2 | 129 | 71 | 2 | 43 | 35
Participants | 97 | 31 | 19 | 0 | 0 | 0 | 14 | 0 | 2 | 0 | 0 | 2 | 2

2. Primary Outcome: Number of Participants With Infusion-related Reactions (Ph1, Ph2, Ph3 Cohort 1 - Cohort 3)
Description: Primary:
  Phase 1, Phase 3 (Cohort 2 and Cohort 3)
  Secondary:
  Phase 2, Phase 3 (Cohort 1)
Time Frame: Through Day 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Combined Phases 1, 2, & 3 Cohort 1 Symptomatic (2.4g IV): Pooled analysis of Phases 1, 2, & 3 Cohort 1 Symptomatic Participants for dosage of 2.4g IV
- Combined Phases 1,2, & 3 Cohort 1 Symptomatic (8.0g IV): Pooled analysis of Phases 1, 2, & 3 Cohort 1 Symptomatic Participants for dosage of 8.0g IV
- Phase 3 Cohort 1 (1.2g IV) Symptomatic: Phase 3 Cohort 1 Symptomatic Participants for dosage of 1.2g IV
Arm/Group | Combined Phases 1, 2, & 3 Cohort 1 Symptomatic (Placebo) | Combined Phases 1, 2, & 3 Cohort 1 Symptomatic (2.4g IV) | Combined Phases 1,2, & 3 Cohort 1 Symptomatic (8.0g IV) | Phase 2 Asymptomatic (Placebo) | Phase 2 Asymptomatic (2.4g IV) | Phase 2 Asymptomatic (8.0g IV) | Phase 3 Cohort 1 (1.2g IV) Symptomatic | Phase 3 Cohort 2 Pediatric (Placebo) | Phase 3 Cohort 2 Pediatric (1.2g IV) | Phase 3 Cohort 2 Pediatric (2.4g IV) | Phase 3 Cohort 3 Pregnant (Placebo) | Phase 3 Cohort 3 Pregnant (1.2g IV) | Phase 3 Cohort 3 Pregnant (2.4g IV)
Number analyzed (Participants) | 2609 | 2614 | 1272 | 74 | 72 | 73 | 1329 | 2 | 129 | 71 | 2 | 43 | 35
Participants | 2 | 4 | 7 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Hypersensitivity Reactions (Ph1, Ph2, Ph3 Cohort 1 - Cohort 3)
Description: Primary:
  Phase 1, Phase 3 (Cohort 2 and Cohort 3)
  Secondary:
  Phase 2, Phase 3 (Cohort 1)
Time Frame: Through Day 29
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Combined Phases 1,2, & 3 Cohort 1 Symptomatic (Placebo): Placebo of R10933 + R10987 Adult Symptomatic Participants with COVID-19
- Combined Phases 1,2, & 3 Cohort 1 Symptomatic (8.0g IV): 8.0g of R10933 + R10987 Adult Symptomatic Participants with COVID-19
Arm/Group | Combined Phases 1,2, & 3 Cohort 1 Symptomatic (Placebo) | Combined Phases 1, 2, & 3 Cohort 1 Symptomatic (2.4g IV) | Combined Phases 1,2, & 3 Cohort 1 Symptomatic (8.0g IV) | Phase 2 Asymptomatic (Placebo) | Phase 2 Asymptomatic (2.4g IV) | Phase 2 Asymptomatic (8.0g IV) | Phase 3 Cohort 1 (1.2g IV) Symptomatic | Phase 3 Cohort 2 Pediatric (Placebo) | Phase 3 Cohort 2 Pediatric (1.2g IV) | Phase 3 Cohort 2 Pediatric (2.4g IV) | Phase 3 Cohort 3 Pregnant (Placebo) | Phase 3 Cohort 3 Pregnant (1.2g IV) | Phase 3 Cohort 3 Pregnant (2.4g IV)
Number analyzed (Participants) | 2609 | 2614 | 1272 | 74 | 72 | 73 | 1329 | 2 | 129 | 71 | 2 | 43 | 35
Participants | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0

4. Primary Outcome: Time-weighted Average Change From Baseline in Viral Load (log10 Copies/mL) From Day 1 to Day 7, as Measured by Quantitative Reverse Transcription Quantitative Polymerase Chain Reaction (RT-qPCR) in Nasopharyngeal (NP) Swab Samples (Ph1, Ph2)
Description: Primary:
  Phase 1, Phase 2
Time Frame: Baseline up to Day 7
Population: All randomized participants in Phase 1 or Phase 2 with qualitatively positive RT-qPCR in NP swab samples at randomization or collected within 2 hours after study drug infusion was initiated. This pooled modified full analysis set (mFAS) includes all randomized patients with positive RT-qPCR in NP swab samples at randomization and is based on the treatment allocated (as randomized).
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- Phase 1 + Phase 2 Symptomatic (Placebo): Pooled Phase 1 + Phase 2 Symptomatic Placebo Participants
- Phase 1 + Phase 2 Symptomatic (2.4g IV): Pooled Phase 1 + Phase 2 Symptomatic 2.4g IV Participants
- Phase 1 + Phase 2 Symptomatic (8.0g IV): Pooled Phase 1 + Phase 2 Symptomatic 8.0g IV Participants
Arm/Group | Phase 1 + Phase 2 Symptomatic (Placebo) | Phase 1 + Phase 2 Symptomatic (2.4g IV) | Phase 1 + Phase 2 Symptomatic (8.0g IV)
Number analyzed (Participants) | 232 | 219 | 220
log10 copies/mL | -1.32 (1.047) | -1.65 (0.977) | -1.67 (1.157)
Statistical Analysis 1: Comparison: Phase 1 + Phase 2 Symptomatic (Placebo) vs Phase 1 + Phase 2 Symptomatic (2.4g IV); Test type: Superiority; p = 0.0006, ANCOVA; LS Mean = -0.33, 95% CI 2-sided [-0.52 to -0.14], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Phase 1 + Phase 2 Symptomatic (Placebo) vs Phase 1 + Phase 2 Symptomatic (8.0g IV); Test type: Superiority; p < 0.0001, ANCOVA; LS Mean = -0.37, 95% CI 2-sided [-0.56 to -0.19], Standard Error of Mean 0.10

5. Primary Outcome: Proportion of Participants With at Least One (≥1) COVID-19-related Hospitalization or All-cause Death (Ph3 Cohort 1- 1.2g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: Participants that were ≥18 years old and not pregnant at randomization, and randomized on or before 17-Jan-2021 with detectable SARS-CoV-2 RNA by RT-qPCR in nasopharyngeal swabs at randomization and at least 1 risk factor for severe COVID-19 at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase 3 Cohort 1 (Placebo) >=18: Phase 3 Cohort 1 (Placebo)
- Phase 3 Cohort 1 (1.2g IV) >= 18: Phase 3 Cohort 1 (1.2g IV)
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Percentage of Participants | 3.2 [2.1 to 4.7] | 1.0 [0.4 to 1.9]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1 (Placebo) >=18 vs Phase 3 Cohort 1 (1.2g IV) >= 18; Test type: Superiority; p = 0.0024, Cochran-Mantel-Haenszel

6. Primary Outcome: Proportion of Participants With at Least One (≥1) COVID-19-related Hospitalization or All-cause Death (Ph3 Cohort 1 - 2.4g vs Placebo)
Description: Primary:
  Phase 3 (Cohort 1)
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase 3 Cohort 1 (2.4g IV) >= 18: Phase 3 Cohort 1 (2.4g IV)
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1341 | 1355
Percentage of Participants | 4.6 [3.6 to 5.9] | 1.3 [0.8 to 2.1]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1 (Placebo) >=18 vs Phase 3 Cohort 1 (2.4g IV) >= 18; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

7. Primary Outcome: Concentration of REGN10983 + REGN10987 in Serum Over Time (Ph3 Cohort 2)
Description: Phase 3 Cohort 2
  [Nominal Sampling Time] = [Clinical Study Time (Visit Day - 1)]
Time Frame: Up to Nominal Sampling Day 28
Population: The pharmacokinetics (PK) analysis population includes all patients who received any study drug (safety population) and who had at least 1 non-missing result following the first dose of study drug
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Phase 3 Cohort 2 Pediatric (1.2g IV) | Phase 3 Cohort 2 Pediatric (2.4g IV)
Number analyzed (Participants) | 129 | 71
mg/L
  Day 0: End of Infusion: number analyzed (Participants) | 107 | 51
  Day 0: End of Infusion | 402 (196) | 710 (275)
  Nominal Sampling Day 28: number analyzed (Participants) | 94 | 48
  Nominal Sampling Day 28 | 108 (60.1) | 198 (78.7)

8. Secondary Outcome: Time to COVID-19 Symptoms Resolution (Ph3 Cohort 1 - 1.2g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Up to Day 29
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Phase 3 Cohort 1 (Placebo): Phase 3 Cohort 1 (Placebo)
- Phase 3 Cohort 1 (1.2 g IV): Phase 3 Cohort 1 (1.2 g IV) - Post PA6 mFAS
Arm/Group | Phase 3 Cohort 1 (Placebo) | Phase 3 Cohort 1 (1.2 g IV)
Number analyzed (Participants) | 680 | 673
Days | 14.0 [13.0 to 16.0] | 10.0 [9.0 to 12.0]

9. Secondary Outcome: Time to COVID-19 Symptoms Resolution (Ph3 Cohort 1 - 2.4g vs Placebo)
Description: Phase 3 (Cohort 1)
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 3 Age>=18: Placebo | Phase 3 Age>=18: 2.4 IV
Number analyzed (Participants) | 1197 | 1214
Days | 14.0 (13.0) [13.0 to 15.0] | 10.0 (10.0) [10.0 to 11.0]

10. Secondary Outcome: Proportion of Participants With ≥1 COVID-19-related Hospitalization or All-cause Death From Day 4 Through Day 29 (Ph3 Cohort 1 - 1.2g vs. Placebo)
Description: Phase 3 (Cohort 1)
Time Frame: Day 4 thru Day 29
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 735 | 748
Participants | 5 | 18

11. Secondary Outcome: Proportion of Participants With ≥1 COVID-19-related Hospitalization or All-cause Death From Day 4 Through Day 29 (Ph3 Cohort 1 - 2.4g vs. Placebo)
Description: Phase 3 (Cohort 1)
Time Frame: From Day 4 Through Day 29
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1340 | 1351
Participants | 46 | 5

12. Secondary Outcome: Change From Baseline in Viral Load at Each Visit, as Measured by RT-qPCR in Nasopharyngeal Swabs (Next Phase 2 Cohort)
Description: Next Phase 2 Symptomatic
Time Frame: Day 5, Day 7, Day 15, Day 29
Population: Participants analyzed are part of modified Full Analysis Set (mFAS) and have documented status at baseline. Next Phase 2 participants included the next 524 participants randomized to Phase 2 subsequent to the first 275 symptomatic participants randomized in Phase 1 / 2
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Groups:
- Next Phase 2 (Placebo): Next Phase 2 Placebo Participants
- Next Phase 2 (2.4g IV): Next Phase 2 Participants 2.4g IV
- Next Phase 2 (8.0g IV): Next Phase 2 Participants 8.0g IV
Arm/Group | Next Phase 2 (Placebo) | Next Phase 2 (2.4g IV) | Next Phase 2 (8.0g IV)
Number analyzed (Participants) | 151 | 145 | 146
log10 copies/mL
  Day 5: number analyzed (Participants) | 141 | 139 | 137
  Day 5 | -1.79 (0.14) | -2.33 (0.14) | -2.28 (0.14)
  Day 7: number analyzed (Participants) | 141 | 139 | 134
  Day 7 | -2.54 (0.13) | -2.79 (0.13) | -3.08 (0.13)
  Day 15: number analyzed (Participants) | 138 | 140 | 134
  Day 15 | -4.56 (0.14) | -4.67 (0.14) | -4.58 (0.14)
  Day 29: number analyzed (Participants) | 139 | 136 | 140
  Day 29 | -5.42 (0.10) | -5.60 (0.10) | -5.45 (0.10)
Statistical Analysis 1: Comparison: Next Phase 2 (Placebo) vs Next Phase 2 (2.4g IV); Test type: Superiority; p = 0.1903, Mixed Models Analysis
Statistical Analysis 2: Comparison: Next Phase 2 (Placebo) vs Next Phase 2 (8.0g IV); Test type: Superiority; p = 0.8431, Mixed Models Analysis

13. Secondary Outcome: Time-weighted Average Change From Baseline in Viral Load (log10 Copies/mL) From Day 1 to Post-baseline Study Days (Ph1, Ph2)
Description: Phase 1, Phase 2
Time Frame: Day 1 to Day 29
Population: All randomized participants pooled in Phase 1 or Phase 2 with qualitatively positive RT-qPCR in NP swab samples at randomization or collected within 2 hours after study drug infusion was initiated. This modified full analysis set (mFAS) includes all randomized patients with positive RT-qPCR in NP swab samples at randomization and is based on the treatment allocated (as randomized).
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Phase 1 + Phase 2 Symptomatic (Placebo) | Phase 1 + Phase 2 Symptomatic (2.4g IV) | Phase 1 + Phase 2 Symptomatic (8.0g IV)
Number analyzed (Participants) | 232 | 219 | 220
log10 copies/mL
  TWA Change from BL: Day 1 to Day 5: number analyzed (Participants) | 221 | 210 | 213
  TWA Change from BL: Day 1 to Day 5 | -0.93 (0.07) | -1.23 (0.07) | -1.25 (0.07)
  TWA Change from BL: Day 1 to Day 7: number analyzed (Participants) | 224 | 211 | 214
  TWA Change from BL: Day 1 to Day 7 | -1.35 (0.07) | -1.68 (0.08) | -1.72 (0.08)
  TWA Change from BL: Day 1 to Day 15: number analyzed (Participants) | 224 | 212 | 216
  TWA Change from BL: Day 1 to Day 15 | -2.57 (0.07) | -2.93 (0.08) | -2.96 (0.08)
  TWA Change from BL: Day 1 to Day 29: number analyzed (Participants) | 224 | 213 | 216
  TWA Change from BL: Day 1 to Day 29 | -3.74 (0.06) | -3.97 (0.07) | -4.03 (0.07)

14. Secondary Outcome: Percentage of Participants With ≥1 COVID-19-related Medically-attended Visit Through Day 29 (Ph1, Ph2)
Description: Phase 1, Phase 2
Time Frame: Through Day 29
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1 + Phase 2 Symptomatic (Placebo) | Phase 1 + Phase 2 Symptomatic (2.4g IV) | Phase 1 + Phase 2 Symptomatic (8.0g IV)
Number analyzed (Participants) | 232 | 219 | 220
Percentage of Participants | 7.8 [4.7 to 12.0] | 3.2 [1.3 to 6.5] | 2.7 [1.0 to 5.8]

15. Secondary Outcome: Percentage of Participants With ≥1 COVID-19 Related Hospitalization, Emergency Room, or Urgent Care Visit Through Day 29 (Ph1, Ph2)
Description: Phase 1, Phase 2
Time Frame: Through Day 29
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1 + Phase 2 Symptomatic (Placebo) | Phase 1 + Phase 2 Symptomatic (2.4g IV) | Phase 1 + Phase 2 Symptomatic (8.0g IV)
Number analyzed (Participants) | 232 | 219 | 220
Percentage of Participants | 4.7 [2.4 to 8.3] | 2.7 [1.0 to 5.9] | 2.3 [0.7 to 5.2]

16. Secondary Outcome: Time to First Onset of Symptoms Consistent With COVID-19 (Phase 2 Asymptomatic Cohort Only)
Description: Phase 2 Only
Time Frame: Up to Day 29
Population: Phase 2 asymptomatic cohort
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Placebo: Placebo of R10933 + R10987 Adult Participants with asymptomatic SARS-CoV-2 infection
Arm/Group | Placebo | Phase 2 Asymptomatic: 2.4 IV | Phase 2 Asymptomatic: 8.0 IV
Number analyzed (Participants) | 74 | 72 | 73
Days | 4.0 [2.0 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 4.0 [2.0 to NA] — Insufficient number of participants with events

17. Secondary Outcome: Proportion of Participants With ≥1 COVID-19-related Hospitalization, Emergency Room Visit, or All-cause Death (Ph3 Cohort 1) - Placebo vs. 1.2g IV
Description: Phase 3 Cohort 1 - Placebo vs. 1.2 g IV
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Participants | 51 | 20

18. Secondary Outcome: Proportion of Participants With ≥1 COVID-19-related Hospitalization, Emergency Room Visit, or All-cause Death (Ph3 Cohort 1) - Placebo vs. 2.4g IV
Description: Phase 3 (Cohort 1)
Time Frame: Through day 29
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1341 | 1355
Participants | 62 | 18

19. Secondary Outcome: Concentration of REGN10933 + REGN10987 in Serum Over Time (Ph1 Cohort 1, Ph2 Cohort 1, Ph3 Cohort 1 and Cohort 3)
Description: Secondary:
  Phase 1, Phase 2, Phase 3 (Cohort 1 and Cohort 3) - Symptomatic Participants
  [Nominal Sampling Time] = [Clinical Study Time (Visit Day - 1)]
Time Frame: Up to Nominal Sampling Day 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Phase 1 (2.4g IV): Phase 1 (2.4g IV) - PK Analysis Set
- Phase 1 (8.0g IV): Phase 1 (8.0g IV) - PK Analysis Set
- Phase 2 (2.4g IV): Phase 2 (2.4g IV) - PK Analysis Set
- Phase 2 (8.0g IV): Phase 2 (8.0g IV) - PK Analysis Set
- Phase 3 Cohort 1 (1.2g IV): Phase 3 Cohort 1 (1.2g IV) - PK Analysis Set
- Phase 3 Cohort 1 (2.4g IV): Phase 3 Cohort 1 (2.4g IV) - PK Analysis Set
- Phase 3 Cohort 1 (8.0g IV): Phase 3 Cohort 1 (8.0g IV) - PK Analysis Set
- Phase 3 Cohort 3 (1.2g IV): Phase 3 Cohort 3 (1.2g IV) - PK Analysis Set
- Phase 3 Cohort 3 (2.4g IV): Phase 3 Cohort 3 (2.4g IV) - PK Analysis Set
Arm/Group | Phase 1 (2.4g IV) | Phase 1 (8.0g IV) | Phase 2 (2.4g IV) | Phase 2 (8.0g IV) | Phase 3 Cohort 1 (1.2g IV) | Phase 3 Cohort 1 (2.4g IV) | Phase 3 Cohort 1 (8.0g IV) | Phase 3 Cohort 3 (1.2g IV) | Phase 3 Cohort 3 (2.4g IV)
Number analyzed (Participants) | 18 | 20 | 218 | 237 | 3477 | 3477 | 881 | 22 | 37
mg/L
  Day 0: EOI | 594 (276) | 1652 (928) | 701 (287) | 2142 (815) | 415 (178) | 669 (236) | 2239 (740) | 305 (80.8) | 536 (165)
  Day 28 | 141 (97.5) | 384 (143) | 142 (62.5) | 453 (179) | 85.1 (36.9) | 143 (55.1) | 463 (166) | 63.7 (25.9) | 119 (31.1)

20. Secondary Outcome: Assessment of Pharmacokinetic (PK) Parameter: Maximum Serum Concentration Observed (Cmax) of REGN10933+REGN10987 (Phase 1)
Description: Phase 1 Only
Time Frame: Through Day 29
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Phase 1 PK-AS: Phase 1 PK-AS (Pharmacokinetic Analysis Set)
Arm/Group | Phase 1 PK-AS
Number analyzed (Participants) | 45
mg/L
  2.4g IV: number analyzed (Participants) | 22
  2.4g IV | 689 (391)
  8.0g IV: number analyzed (Participants) | 23
  8.0g IV | 1805 (720)

21. Secondary Outcome: Assessment of PK Parameter: Time to Cmax (Tmax) for REGN10933+REGN10987 (Phase 1)
Description: Phase 1 Only
Time Frame: Through Day 29
Population: as for outcome 7
Measure: Median (Full Range); unit: Days
Arm/Group | Phase 1 PK-AS
Number analyzed (Participants) | 45
Days
  2.4g IV: number analyzed (Participants) | 22
  2.4g IV | 27.7 [0.0847 to 28.2]
  8.0g IV: number analyzed (Participants) | 23
  8.0g IV | 0.0854 [0.0431 to 2.06]

22. Secondary Outcome: Assessment of PK Parameter: Area Under the Curve (AUC) Computed From Time Zero to Day 28 Concentration (AUC 0-28) for REGN10933+REGN10987 (Phase 1)
Description: Phase 1 Only
Time Frame: Through Day 29
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: day*milligram/Liter
Arm/Group | Phase 1 PK-AS
Number analyzed (Participants) | 45
day*milligram/Liter
  2.4g IV: number analyzed (Participants) | 19
  2.4g IV | 7158 (4255)
  8.0g IV: number analyzed (Participants) | 20
  8.0g IV | 19084 (5172)

23. Secondary Outcome: Immunogenicity as Measured by Anti-drug (ADA) to REGN10933 (Ph1 Cohort 1, Ph2 Cohort 1, Ph3 Cohort 1)
Description: Phase 1, Phase 2, Phase 3 (Cohort 1) - Pooled Symptomatic Participants
Time Frame: Through Day 29
Population: The anti-drug antibody (ADA) analysis set (AAS) includes all subjects who received any study drug (safety population) and had at least one non-missing ADA result from the ADA assay after first dose of the study drug(s). Pooled participants will be analyzed according to the treatment actually received. This is an adaptive master protocol design, to allow for flexible adaptation for participants with symptomatic COVID-19, as well as with those with asymptomatic SARS-CoV-2.
Measure: Number; unit: Participants
Groups:
- Phases 1,2, & 3 Cohort 1 Symptomatic (Placebo): Pooled analysis of Phases 1, 2, & 3 Cohort 1 Symptomatic Participants for Placebo
- Phases 3 Cohort 1 Symptomatic (1.2g IV): Phase 3 Cohort 1 Symptomatic Participants for dosage of 1.2g IV
- Phases 1, 2, & 3 Cohort 1 Symptomatic (2.4g IV): Pooled analysis of Phases 1, 2, & 3 Cohort 1 Symptomatic Participants for dosage of 2.4g IV
- Phases 1,2, & 3 Cohort 1 Symptomatic (8.0g IV): Pooled analysis of Phases 1, 2, & 3 Cohort 1 Symptomatic Participants for dosage of 8.0g IV
Arm/Group | Phases 1,2, & 3 Cohort 1 Symptomatic (Placebo) | Phases 3 Cohort 1 Symptomatic (1.2g IV) | Phases 1, 2, & 3 Cohort 1 Symptomatic (2.4g IV) | Phases 1,2, & 3 Cohort 1 Symptomatic (8.0g IV)
Number analyzed (Participants) | 2609 | 1935 | 3087 | 1272
Participants | 17 | 29 | 20 | 1

24. Secondary Outcome: Immunogenicity as Measured by Anti-drug (ADA) to REGN10933 (Ph3 Cohort 2 - Cohort 3)
Description: Symptomatic Participants Phase 3 Cohort 2 Participants Phase 3 Cohort 3 Participants
Time Frame: Through Day 29
Population: The anti-drug antibody (ADA) analysis set (AAS) includes all subjects who received any study drug (safety population) and had at least one non-missing ADA result from the ADA assay after first dose of the study drug(s). Participants will be analyzed according to the treatment actually received. This is an adaptive master protocol design, to allow for flexible adaptation for participants with symptomatic COVID-19, as well as with those with asymptomatic SARS-CoV-2.
Measure: Number; unit: Participants
Groups:
- Phase 3 Cohort 2 (Placebo): Phase 3 Cohort 2 (Placebo) - ADA Analysis Set
- Phase 3 Cohort 2 (1.2g IV): Phase 3 Cohort 2 (1.2g IV) - ADA Analysis Set
- Phase 3 Cohort 2 (2.4g IV): Phase 3 Cohort 2 (2.4g IV) - ADA Analysis Set
- Phase 3 Cohort 3 (Placebo): Phase 3 Cohort 3 (Placebo) - ADA Analysis Set
- Phase 3 Cohort 3 (1.2g IV): Phase 3 Cohort 3 (1.2g IV) - ADA Analysis Set
- Phase 3 Cohort 3 (2.4g IV): Phase 3 Cohort 3 (2.4g IV) - ADA Analysis Set
Arm/Group | Phase 3 Cohort 2 (Placebo) | Phase 3 Cohort 2 (1.2g IV) | Phase 3 Cohort 2 (2.4g IV) | Phase 3 Cohort 3 (Placebo) | Phase 3 Cohort 3 (1.2g IV) | Phase 3 Cohort 3 (2.4g IV)
Number analyzed (Participants) | 1 | 123 | 64 | 1 | 39 | 33
Participants | 0 | 1 | 0 | 0 | 0 | 1

25. Secondary Outcome: Immunogenicity as Measured by ADA to REGN10987 (Ph1 Cohort 1, Ph2 Cohort 1, Ph3 Cohort 1)
Description: Phase 1, Phase 2, Phase 3 (Cohort 1) - Pooled Symptomatic Participants
Time Frame: Through Day 29
Population: as for outcome 23
Measure: Number; unit: Participants
Groups:
- Pooled Phases 1,2, & 3 Cohort 1 Symptomatic (Placebo): Pooled analysis of Phases 1, 2, & 3 Cohort 1 Symptomatic Participants for Placebo
- Phase 3 Cohort 1 Symptomatic (1.2g IV): Phases 3 Cohort 1 Symptomatic Participants for dosage of 1.2g IV
- Pooled Phases 1, 2, & 3 Cohort 1 Symptomatic (2.4g IV): Pooled analysis of Phases 1, 2, & 3 Cohort 1 Symptomatic Participants for dosage of 2.4g IV
- Pooled Phases 1,2, & 3 Cohort 1 Symptomatic (8.0g IV): Pooled analysis of Phases 1, 2, & 3 Cohort 1 Symptomatic Participants for dosage of 8.0g IV
Arm/Group | Pooled Phases 1,2, & 3 Cohort 1 Symptomatic (Placebo) | Phase 3 Cohort 1 Symptomatic (1.2g IV) | Pooled Phases 1, 2, & 3 Cohort 1 Symptomatic (2.4g IV) | Pooled Phases 1,2, & 3 Cohort 1 Symptomatic (8.0g IV)
Number analyzed (Participants) | 2609 | 1934 | 3084 | 1272
Participants | 59 | 56 | 54 | 2

26. Secondary Outcome: Immunogenicity as Measured by ADA to REGN10987 (Ph3 Cohort 2 and Cohort 3)
Description: Symptomatic Participants Phase 3 Cohort 2 Participants Phase 3 Cohort 3 Participants
Time Frame: Through Day 29
Population: as for outcome 24
Measure: Number; unit: Participants
Groups:
- Phase 3 Cohort 2 (Placebo): Phase 3 Cohort 2 Pediatric (Placebo)
- Phase 3 Cohort 2 (1.2g IV): Phase 3 Cohort 2 Pediatric (1.2g IV)
- Phase 3 Cohort 2 (2.4g IV): Phase 3 Cohort 2 Pediatric (2.4g IV)
- Phase 3 Cohort 3 (Placebo): Phase 3 Cohort 3 Pregnant (Placebo)
- Phase 3 Cohort 3 (1.2g IV): Phase 3 Cohort 3 Pregnant (1.2g IV)
- Phase 3 Cohort 3 (2.4g IV): Phase 3 Cohort 3 Pregnant (2.4g IV)
Arm/Group | Phase 3 Cohort 2 (Placebo) | Phase 3 Cohort 2 (1.2g IV) | Phase 3 Cohort 2 (2.4g IV) | Phase 3 Cohort 3 (Placebo) | Phase 3 Cohort 3 (1.2g IV) | Phase 3 Cohort 3 (2.4g IV)
Number analyzed (Participants) | 1 | 123 | 64 | 1 | 39 | 33
Participants | 0 | 1 | 0 | 0 | 2 | 1

27. Secondary Outcome: Immunogenicity as Measured by Neutralizing Antibodies (NAbs) to REGN10933 (Ph3 Cohort 2, Ph3 Cohort 3)
Description: Symptomatic Participants Phase 3 Cohort 2 Participants Phase 3 Cohort 3 Participants
  (TE&TB+;NAb+) = TE = Treatment-emergent; TB = Treatment-boosted; NAb+ = Positive in NAb assay
Time Frame: Through Day 29
Population: as for outcome 24
Measure: Number; unit: Participants
Arm/Group | Phase 3 Cohort 2 (Placebo) | Phase 3 Cohort 2 (1.2g IV) | Phase 3 Cohort 2 (2.4g IV) | Phase 3 Cohort 3 (Placebo) | Phase 3 Cohort 3 (1.2g IV) | Phase 3 Cohort 3 (2.4g IV)
Number analyzed (Participants) | 1 | 123 | 64 | 1 | 39 | 33
Participants | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Immunogenicity as Measured by NAbs to REGN10987 (Ph3 Cohort 2 - Cohort 3)
Description: Phase 3 Cohort 2 Participants Phase 3 Cohort 3 Participants
  (TE&TB+;NAb+) = TE = Treatment-emergent; TB = Treatment-boosted; NAb+ = Positive in NAb assay
Time Frame: Through Day 29
Population: The anti-drug antibody (ADA) analysis set (AAS) includes all subjects who received any study drug (safety population) and had at least one non-missing ADA result from the ADA assay after first dose of the study drug(s). Participants will be analyzed according to the treatment actually received.
Measure: Number; unit: Participants
Arm/Group | Phase 3 Cohort 2 (Placebo) | Phase 3 Cohort 2 (1.2g IV) | Phase 3 Cohort 2 (2.4g IV) | Phase 3 Cohort 3 (Placebo) | Phase 3 Cohort 3 (1.2g IV) | Phase 3 Cohort 3 (2.4g IV)
Number analyzed (Participants) | 1 | 123 | 64 | 1 | 39 | 33
Participants | 0 | 1 | 0 | 00 | 0 | 0

29. Secondary Outcome: Number of Participants With at Least One (≥1) COVID-19-related Hospitalization or All-cause Death (Phase 3 Cohort 2)
Description: Phase 3 (Cohort 2)
Time Frame: Through Day 29
Population: Participants <18 years old who, at baseline, were not pregnant, had symptomatic COVID-19, and had at least 1 risk factor for developing severe disease
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3 Cohort 2 Pediatric (Placebo) | Phase 3 Cohort 2 Pediatric (1.2g IV) | Phase 3 Cohort 2 Pediatric (2.4g IV)
Number analyzed (Participants) | 1 | 121 | 70
Participants | 0 | 0 | 0

30. Secondary Outcome: Percentage of Participants With ≥1 COVID-19-related Medically-attended Visit (Phase 1, Phase 2)
Description: Phase 1, Phase 2 Medically-attended Visits include Hospitalizations, ER visits, Urgent Care Clinic visits, Outpatient/physician office/telemedicine visits
Time Frame: Through Day 29
Population: All randomized participants in Phase 1 or Phase 2 with qualitatively positive RT-qPCR in NP swab samples at randomization or collected within 2 hours after study drug infusion was initiated. This modified full analysis set (mFAS) includes all randomized patients with positive RT-qPCR in NP swab samples at randomization and is based on the treatment allocated (as randomized).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1 + Phase 2 Symptomatic (Placebo) | Phase 1 + Phase 2 Symptomatic (2.4g IV) | Phase 1 + Phase 2 Symptomatic (8.0g IV)
Number analyzed (Participants) | 232 | 219 | 220
Percentage of Participants | 7.8 [4.7 to 12.0] | 3.2 [1.3 to 6.5] | 2.7 [1.0 to 5.8]

31. Secondary Outcome: Percentage of Participants With ≥2 COVID-19-related Medically-attended Visit - (Ph3 Cohort 1) - Placebo vs. 1.2g IV
Description: Phase 3 (Cohort 1)
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase 3 Cohort 1 (Placebo): Phase 3 Cohort 1 (Placebo) Participants
- Phase 3 Cohort 1 (1.2g IV) >=18: Phase 3 Cohort 1 (1.2g IV) Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) | Phase 3 Cohort 1 (1.2g IV) >=18
Number analyzed (Participants) | 748 | 736
Percentage of Participants | 0.5 [0.1 to 1.4] | 0.4 [0.1 to 1.2]

32. Secondary Outcome: Percentage of Participants With ≥2 COVID-19-related Medically-attended Visit - (Ph3 Cohort 1) - Placebo vs. 2.4g IV
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase 3 Cohort 1 (2.4g IV) >=18: Phase 3 Cohort 1 (2.4g IV) Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) | Phase 3 Cohort 1 (2.4g IV) >=18
Number analyzed (Participants) | 1341 | 1355
Percentage of Participants | 1.1 [0.6 to 1.8] | 0.07 [0.0 to 0.4]

33. Secondary Outcome: Total Number of COVID-19-related Medically-attended Visits (Phase 1 and Phase 2)
Description: Phase 1 and Phase 2
Time Frame: Through Day 29
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Groups:
- Phase 1 + Phase 2 Symptomatic: Pooled Phase 1 + Phase 2 Symptomatic Participants mFAS (modified Full Analysis Set)
- Phase 1 + Phase 2 Symptomatic 2.4g IV: Pooled Phase 1 + Phase 2 Symptomatic 2.4g IV mFAS (modified Full Analysis Set)
- Phase 1 + Phase 2 Symptomatic 8.0g IV mFAS (Modified Full Analysis Set): Pooled Phase 1 + Phase 2 Symptomatic 8.0g IV mFAS (modified Full Analysis Set)
Arm/Group | Phase 1 + Phase 2 Symptomatic | Phase 1 + Phase 2 Symptomatic 2.4g IV | Phase 1 + Phase 2 Symptomatic 8.0g IV mFAS (Modified Full Analysis Set)
Number analyzed (Participants) | 232 | 219 | 220
Number of Participants | 18 | 7 | 6

34. Secondary Outcome: Assessment of Pharmacokinetic (PK) Parameter: Maximum Serum Concentration Observed (Cmax) of REGN10933 and REGN10987 (Phase 1 Only)
Description: Phase 1 Only
Time Frame: Through Day 29
Population: The pharmacokinetics (PK) analysis pooled population includes all patients who received any study drug (safety population) and who had at least 1 non-missing result following the first dose of study drug
Measure: Mean (Standard Deviation); unit: mg/L (milligram/Liters)
Groups:
- Phase 1 PK-AS (Pharmacokinetic Analysis Analysis Set): PK-AS of participants in Phase 1 Adult Symptomatic Participants with COVID-19
Arm/Group | Phase 1 PK-AS (Pharmacokinetic Analysis Analysis Set)
Number analyzed (Participants) | 45
mg/L (milligram/Liters)
  REGN10933: number analyzed (Participants) | 22
  REGN10933 | 343 (160)
  REGN10987: number analyzed (Participants) | 22
  REGN10987 | 353 (233)

35. Secondary Outcome: Assessment of PK Parameter: Cmax-to-dose Ratio (Cmax/Dose) of REGN10933 and REGN10987 (Phase 1 Only)
Description: Phase 1 Only
Time Frame: Though Day 29
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/L/mg (milligram/Liter/milligram)
Arm/Group | Phase 1 PK-AS (Pharmacokinetic Analysis Analysis Set)
Number analyzed (Participants) | 45
mg/L/mg (milligram/Liter/milligram)
  REGN10933: number analyzed (Participants) | 22
  REGN10933 | 0.286 (0.134)
  REGN10987: number analyzed (Participants) | 22
  REGN10987 | 0.294 (0.194)

36. Secondary Outcome: Assessment of PK Parameter: Time to Cmax (Tmax) for REGN10933 and REGN10987 (Phase 1 Only)
Description: Phase 1 Only
Time Frame: Through Day 29
Population: as for outcome 7
Measure: Median (Full Range); unit: Day
Arm/Group | Phase 1 PK-AS (Pharmacokinetic Analysis Analysis Set)
Number analyzed (Participants) | 45
Day
  REGN10933: number analyzed (Participants) | 22
  REGN10933 | 0.0861 [0 to 14.9]
  REGN10987: number analyzed (Participants) | 22
  REGN10987 | 0.0861 [0 to 14.9]

37. Secondary Outcome: Assessment of PK Parameter: Area Under the Curve (AUC) Computed From Time Zero to the Time of the Last Positive Concentration (AUClast) for REGN10933 - (Phase 1 Only)
Description: Phase 1 Only - Tlast (Time of last quantifiable concentration)
Time Frame: Through Day 29
Population: as for outcome 7
Measure: Median (Full Range); unit: ((day*mg/L)/mg)
Groups:
- Phase 1 PK-AS (Pharmacokinetic Analysis Set): PK-AS of participants in Phase 1 Adult Symptomatic Participants with COVID-19
Arm/Group | Phase 1 PK-AS (Pharmacokinetic Analysis Set)
Number analyzed (Participants) | 22
((day*mg/L)/mg)
  REGN10933 | 27.7 [0.0847 to 28.2]
  REGN10987 | 27.7 [13.0 to 28.2]

38. Secondary Outcome: Proportion of Participants With at Least One (≥1) COVID-19-related Hospitalization or All-cause Death From Day 4 Through Day 29 (Ph3 Cohort 1- 1.2g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Day 4 Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Percentage of Participants | 2.4 [1.4 to 3.8] | 0.7 [0.2 to 1.6]

39. Secondary Outcome: Proportion of Participants With at Least One (≥1) COVID-19-related Hospitalization or All-cause Death From Day 4 Through Day 29 (Ph3 Cohort 1- 2.4g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Day 4 Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1340 | 1351
Percentage of Participants | 3.4 [2.5 to 4.6] | 0.4 [0.1 to 0.9]

40. Secondary Outcome: Proportion of Participants With at Least One (≥1) COVID-19-related Medically-attended Visit or All-cause Death Through Day 29 (Ph3 Cohort 1- 1.2g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Percentage of Participants | 6.8 [5.1 to 8.9] | 2.7 [1.7 to 4.2]

41. Secondary Outcome: Proportion of Participants With at Least One (≥1) COVID-19-related Medically-attended Visit or All-cause Death Through Day 29 (Ph3 Cohort 1- 2.4g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1341 | 1355
Percentage of Participants | 8.1 [6.7 to 9.7] | 3.2 [2.3 to 4.3]

42. Secondary Outcome: Number of Participants With at Least One (≥1) COVID-19-related Medically-attended Visit or All-cause Death Through Day 29 (Phase 3 Cohort 2)
Description: Phase 3 (Cohort 2)
Time Frame: Through Day 29
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3 Cohort 2 Pediatric (Placebo) | Phase 3 Cohort 2 Pediatric (1.2g IV) | Phase 3 Cohort 2 Pediatric (2.4g IV)
Number analyzed (Participants) | 1 | 121 | 70
Participants | 0 | 2 | 1

43. Secondary Outcome: Proportion of Participants With at Least One (≥1) COVID-19-related Medically-attended Visit by Type of Visit Through Day 29 (Ph3 Cohort 1- 1.2g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Percentage of Participants
  Hospitalization | 3.1 [2.0 to 4.6] | 0.8 [0.3 to 1.8]
  Emergency Room | 1.3 [0.6 to 2.4] | 0.3 [0.0 to 1.0]
  Urgent Care | 0.7 [0.2 to 1.6] | 0.1 [0.0 to 0.8]
  Physician office visit/Telemedicine | 1.6 [0.8 to 2.8] | 1.4 [0.7 to 2.5]

44. Secondary Outcome: Proportion of Participants With at Least One (≥1) COVID-19-related Medically-attended Visit by Type of Visit Through Day 29 (Ph3 Cohort 1- 2.4g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1341 | 1355
Percentage of Participants
  Hospitalization | 4.4 [3.4 to 5.6] | 1.3 [0.7 to 2.0]
  Emergency Room | 1.2 [0.7 to 1.9] | 0.7 [0.3 to 1.3]
  Urgent Care | 0.5 [0.2 to 1.1] | 0.2 [0.0 to 0.6]
  Physician office visit/Telemedicine | 1.8 [1.1 to 2.7] | 1.0 [0.5 to 1.6]

45. Secondary Outcome: Total Number of COVID-19-related Medically-attended Visits by Type of Visit Through Day 29 (Phase 3 Cohort 2)
Description: Phase 3 (Cohort 2)
Time Frame: Through Day 29
Population: as for outcome 29
Measure: Number; unit: Medically-Attended Visit
Arm/Group | Phase 3 Cohort 2 Pediatric (Placebo) | Phase 3 Cohort 2 Pediatric (1.2g IV) | Phase 3 Cohort 2 Pediatric (2.4g IV)
Number analyzed (Participants) | 1 | 121 | 70
Medically-Attended Visit
  Emergency Room | 0 | 1 | 0
  Outpatient/Telemedicine | 0 | 1 | 1

46. Secondary Outcome: Cumulative Incidence Percentage of Patients With COVID-19-related Hospitalization or All-cause Death Through Day 29 (Ph3 Cohort 1- 1.2g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Cumulative Incidence Percentage | 3.2 [2.2 to 4.8] | 1.0 [0.5 to 2.0]

47. Secondary Outcome: Cumulative Incidence Percentage of Patients With COVID-19-related Hospitalization or All-cause Death Through Day 29 (Ph3 Cohort 1- 2.4g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1341 | 1355
Cumulative Incidence Percentage | 4.6 [3.6 to 5.9] | 1.3 [0.8 to 2.1]

48. Secondary Outcome: Cumulative Incidence Percentage of Patients With COVID-19-related Hospitalization, Emergency Room (ER) or All-cause Death Through Day 29 (Ph3 Cohort 1- 1.2g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Cumulative Incidence Percentage | 4.6 [3.3 to 6.3] | 1.2 [0.6 to 2.4]

49. Secondary Outcome: Cumulative Incidence Percentage of Patients With COVID-19-related Hospitalization, Emergency Room (ER) or All-cause Death Through Day 29 (Ph3 Cohort 1- 2.4g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1341 | 1355
Cumulative Incidence Percentage | 5.8 [4.7 to 7.2] | 2.0 [1.4 to 2.9]

50. Secondary Outcome: Cumulative Incidence Percentage of Patients With COVID-19-related Medically-attended Visit or All-cause Death Through Day 29 (Ph3 Cohort 1- 1.2g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Cumulative Incidence Percentage | 6.9 [5.2 to 8.9] | 2.7 [1.8 to 4.2]

51. Secondary Outcome: Cumulative Incidence Percentage of Patients With COVID-19-related Medically-attended Visit or All-cause Death Through Day 29 (Ph3 Cohort 1- 2.4g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1341 | 1355
Cumulative Incidence Percentage | 8.2 [6.8 to 9.8] | 3.2 [2.4 to 4.3]

52. Secondary Outcome: Proportion of Participants Requiring Supplemental Oxygen Due to COVID-19 by Day 29 (Ph3 Cohort 1- 1.2g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Percentage of Participants | 2.1 [1.2 to 3.5] | 0.5 [0.1 to 1.4]

53. Secondary Outcome: Proportion of Participants Requiring Supplemental Oxygen Due to COVID-19 by Day 29 (Ph3 Cohort 1- 2.4g vs Placebo)
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1341 | 1355
Percentage of Participants | 3.6 [2.7 to 4.7] | 1.0 [0.5 to 1.6]

54. Secondary Outcome: Percentage of Participants With All-Cause Death (Ph3 Cohort 1) Placebo vs. 1.2g
Description: Phase 3 Cohort 1
Time Frame: by Day 29, Day 120, and Day 169
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Percentage of Participants
  by Day 29 | 0.1 [0.0 to 0.7] | 0.1 [0.0 to 0.8]
  by Day 120 | 0.1 [0.0 to 0.7] | 0.1 [0.0 to 0.8]
  by Day 169 | 0.1 [0.0 to 0.7] | 0.1 [0.0 to 0.8]

55. Secondary Outcome: Percentage of Participants With All-Cause Death (Ph3 Cohort 1) Placebo vs. 2.4g
Description: Phase 3 Cohort 1 Placebo vs. 2.4g IV
Time Frame: by Day 29, Day 120, and Day 169
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >=18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1341 | 1355
Percentage of Participants
  by Day 29 | 0.2 [0.0 to 0.7] | 0.07 [0.0 to 0.4]
  by Day 120 | 0.4 [0.1 to 0.9] | 0.07 [0.0 to 0.4]
  by Day 169 | 0.1 [0.1 to 0.9] | 0.07 [0.0 to 0.4]

56. Secondary Outcome: Proportion of Participants With High Viral Load at Each Visit - (Phase 2 Only)
Description: Next Phase 2 Only
Time Frame: Through Day 29
Population: In light of evolving information concerning SARS-CoV-2 infection, including the profile of viral load among patients and the adequacy of sampling methodologies, virologic efficacy endpoints and sampling methods were modified during the course of the study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Placebo: Placebo Phase 2 Participants
- R10933+R10987 2.4 g IV: R10933+R10987 2.4 g IV
- R10933+R10987 8.0 g IV: R10933+R10987 8.0 g IV
Arm/Group | Placebo | R10933+R10987 2.4 g IV | R10933+R10987 8.0 g IV
Number analyzed (Participants) | 150 | 142 | 145
Percentage of Participants
  Day 3: number analyzed (Participants) | 136 | 132 | 135
  Day 3 | 77.2 [69.2 to 84.0] | 67.4 [58.7 to 75.3] | 62.2 [53.5 to 70.4]
  Day 5: number analyzed (Participants) | 140 | 134 | 136
  Day 5 | 61.4 [52.8 to 69.5] | 47.0 [38.3 to 55.8] | 44.1 [35.6 to 52.9]
  Day 7: number analyzed (Participants) | 139 | 131 | 132
  Day 7 | 48.9 [40.4 to 57.5] | 31.3 [23.5 to 40.0] | 28.8 [21.2 to 37.2]
  Day 15: number analyzed (Participants) | 100 | 98 | 95
  Day 15 | 10.0 [4.9 to 17.6] | 5.1 [1.7 to 11.5] | 4.2 [1.2 to 10.4]
  Day 29: number analyzed (Participants) | 53 | 49 | 55
  Day 29 | 0 [0 to 0] | 2.0 [0.1 to 10.9] | 1.8 [0.0 to 9.7]

57. Secondary Outcome: Correlation of RT-qPCR Results Over Time Between Different Sample Types (NP, Nasal, and Saliva) - (Phase 1 Only)
Description: Phase 1 Only
Time Frame: Up to Day 29
Population: Nasal and saliva sample collection was discontinued early in the study because nasopharyngeal samples were determined to be more reliable for quantitative analysis. Therefore, data was not collected for this outcome measure. The Phase 1/2 SAP does not specify any analyses related to nasal and saliva samples collections
Groups:
- Phase 1 Only: Phase 1 Only Participants
Arm/Group | Phase 1 Only
Number analyzed (Participants) | 0

58. Secondary Outcome: Change From Baseline in Viral Load at Each Visit, as Measured by RT-qPCR in Nasal Swabs - (Phase 1 Only)
Description: Phase 1 Only
Time Frame: Baseline Up To Day 29
Population: as for outcome 57
Groups:
- Phase 1 Only: Phase 1 Participants
Arm/Group | Phase 1 Only
Number analyzed (Participants) | 0

59. Secondary Outcome: Change From Baseline in Viral Load at Each Visit, as Measured by RT-qPCR in Saliva Samples - (Phase 1 Only)
Description: Phase 1 Only
Time Frame: Baseline Up to Day 29
Population: as for outcome 57
Groups:
- Phase 1: Adult Symptomatic Participants with COVID-19
Arm/Group | Phase 1
Number analyzed (Participants) | 0

60. Secondary Outcome: Concordance of RT-qPCR Results Over Time Between Different Sample Types (NP, Nasal, and Saliva) - (Phase 1 Only)
Description: Phase 1 Only
Time Frame: Up To Day 29
Population: as for outcome 57
Groups:
- Phase 1 Only: Phase 1 Participants Only
Arm/Group | Phase 1 Only
Number analyzed (Participants) | 0

61. Secondary Outcome: Time-weighted Average Change From Baseline in Viral Load (log10 Copies/mL), as Measured by RT-qPCR in Saliva Samples - (Phase 1)
Description: Phase 1 Only
Time Frame: Baseline up to Day 22
Population: as for outcome 56
Groups:
- Phase 1: Phase 1 Participants
Arm/Group | Phase 1
Number analyzed (Participants) | 0

62. Secondary Outcome: Number of Participants With Viral Loads Below the Limit of Detection at Each Visit - (Phase 2 Only)
Description: Phase 2 Only
Time Frame: Through Day 29
Population: as for outcome 56
Measure: Number; unit: Number of Participants
Groups:
- Phase 2 Only (Placebo): Phase 2 (Placebo) Asymptomatic Participants
- Phase 2 (2.4g IV) Participants: Phase 2 (2.4 g IV) Asymptomatic Participants of modified Full Analysis Set (mFAS)
- Phase 2 (8.0g IV) Participants: Phase 2 (8.0g IV) Asymptomatic Participants of modified Full Analysis Set (mFAS)
Arm/Group | Phase 2 Only (Placebo) | Phase 2 (2.4g IV) Participants | Phase 2 (8.0g IV) Participants
Number analyzed (Participants) | 57 | 49 | 51
Number of Participants
  Day 0 (Baseline) | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 54 | 45 | 47
  Day 5 | 14 | 15 | 10
  Day 7: number analyzed (Participants) | 55 | 48 | 48
  Day 7 | 18 | 22 | 14
  Day 15: number analyzed (Participants) | 56 | 47 | 50
  Day 15 | 36 | 39 | 32
  Day 29: number analyzed (Participants) | 54 | 46 | 46
  Day 29 | 48 | 44 | 36

63. Secondary Outcome: Duration of Symptoms Consistent With COVID-19 (Phase 2 Only)
Description: Phase 2 Only
Time Frame: Through Day 29
Population: Participants who were part of Phase 2 Asymptomatic modified Full Analysis Set (mFAS)
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Phase 2 Placebo: Phase 2 (Placebo) Asymptomatic Participants
- Phase 2 (2.4 g IV) Participants: Phase 2 (2.4 g IV) Asymptomatic Participants of modified Full Analysis Set (mFAS)
Arm/Group | Phase 2 Placebo | Phase 2 (2.4 g IV) Participants | Phase 2 (8.0g IV) Participants
Number analyzed (Participants) | 22 | 14 | 17
Days | 12.6 (9.27) | 13.1 (9.34) | 14.4 (10.95)

64. Secondary Outcome: Time to First Onset of Symptoms Consistent With COVID-19 (Phase 2 Asymptomatic Cohort Only)
Description: Phase 2 Only
Time Frame: Through Day 29
Population: Phase 2 asymptomatic cohort
Measure: Median (Full Range); unit: Days
Groups:
- Phase 2 Only: Phase 2 Participants
- Phase 2 2.4g IV: Phase 2 asymptomatic participants
- Phase 2 8.0g IV: Phase 2 asymptomatic participants 8.0g IV
Arm/Group | Phase 2 Only | Phase 2 2.4g IV | Phase 2 8.0g IV
Number analyzed (Participants) | 57 | 49 | 51
Days | 3.0 [1.0 to 9.0] | 2.5 [1.0 to NA] — Inadequate number of events to reach upper limit | 4.0 [2.0 to NA] — Inadequate number of events to reach upper limit

65. Secondary Outcome: Number of Participants Admitted to a Hospital Due to COVID-19 (Phase 1, Phase 2)
Description: Phase 1, Phase 2
Time Frame: Through Day 29
Population: All pooled randomized participants in Phase 1 or Phase 2 with qualitatively positive RT-qPCR in NP swab samples at randomization or collected within 2 hours after study drug infusion was initiated. This modified full analysis set (mFAS) includes all randomized patients with positive RT-qPCR in NP swab samples at randomization and is based on the treatment allocated (as randomized).
Measure: Number (95% Confidence Interval); unit: Number Participants
Groups:
- Phase 1 + Phase 2 Symptomatic (Placebo) Participants: Pooled Phase 1 + Phase 2 Symptomatic Placebo Participants
- Phase 1 + Phase 2 Symptomatic (2.4g IV) Participants: Pooled Phase 1 + Phase 2 Symptomatic (2.4g IV) Participants
- Phase 1 + Phase 2 Symptomatic (8.0g IV) Participants: Pooled Phase 1 + Phase 2 Symptomatic (8.0g IV) Participants
Arm/Group | Phase 1 + Phase 2 Symptomatic (Placebo) Participants | Phase 1 + Phase 2 Symptomatic (2.4g IV) Participants | Phase 1 + Phase 2 Symptomatic (8.0g IV) Participants
Number analyzed (Participants) | 81 | 73 | 74
Number Participants | 1 [0.0 to 6.7] | 0 [0 to 0] | 0 [0 to 0]

66. Secondary Outcome: Time to Negative RT-qPCR in All Tested Samples With no Subsequent Positive RT-qPCR in Any Tested Samples - (Phase 1 Only)
Description: Phase 1 Only
Time Frame: Through Day 29
Population: as for outcome 56
Arm/Group | Phase 1 Only
Number analyzed (Participants) | 0

67. Secondary Outcome: Proportion of Participants With All-cause Mortality (Phase 2 Asymptomatic)
Description: Phase 2 Asymptomatic
Time Frame: Through Day 29
Population: Phase 2 asymptomatic cohort
Measure: Number; unit: Participants
Groups:
- Phase 2 Asymptomatic Placebo: Placebo of R10933 + R10987 Adult Participants with asymptomatic SARS-CoV-2 infection
- Phase 2 Asymptomatic R10933+R10987 2.4g IV: 2.4g of R10933 + R10987 Adult Participants with asymptomatic SARS-CoV-2 infection
- Phase 2 Asymptomatic R10933+R10987 8.0g IV: 8.0g of R10933 + R10987 Adult Participants with asymptomatic SARS-CoV-2 infection
Arm/Group | Phase 2 Asymptomatic Placebo | Phase 2 Asymptomatic R10933+R10987 2.4g IV | Phase 2 Asymptomatic R10933+R10987 8.0g IV
Number analyzed (Participants) | 73 | 74 | 75
Participants | 0 | 0 | 0

68. Secondary Outcome: Time to All-cause Death (Ph3 Cohort 1- 1.2g vs Placebo)
Description: Phase 3 Cohort 1 (1.2g IV)
Time Frame: Through Day 169
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Phase 3 Cohort 1 (Placebo) >= 18: Phase 3 Cohort 1 Participants (Placebo)
- Phase 3 Cohort 1 (1.2g IV) >= 18: Phase 3 Cohort 1 Participants (1.2g IV)
Arm/Group | Phase 3 Cohort 1 (Placebo) >= 18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Days | NA [NA to NA] — Unable to calculate due to too few events | NA [NA to NA] — Unable to calculate due to too few events
Statistical Analysis 1: Comparison: Phase 3 Cohort 1 (Placebo) >= 18 vs Phase 3 Cohort 1 (1.2g IV) >= 18; Test type: Superiority; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.06 to 16.12]

69. Secondary Outcome: Time to All-cause Death (Ph3 Cohort 1- 2.4g vs Placebo)
Description: Phase 3 Cohort 1 (2.4g IV)
Time Frame: Through Day 169
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Phase 3 Cohort 1 (2.4g IV) >= 18: Phase 3 Cohort 1 Participants (2.4g IV)
Arm/Group | Phase 3 Cohort 1 (Placebo) >= 18 | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1341 | 1355
Days | NA [NA to NA] — Unable to calculate due to too few events | NA [NA to NA] — Unable to calculate due to too few events
Statistical Analysis 1: Comparison: Phase 3 Cohort 1 (Placebo) >= 18 vs Phase 3 Cohort 1 (2.4g IV) >= 18; Test type: Superiority; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.03 to 3.13]

70. Secondary Outcome: Time to All-cause Death (Phase 3 Cohort 2)
Description: Phase 3 (Cohort 2)
Time Frame: Through Day 29
Population: There were no deaths in this cohort. Phase 3 Cohort 2 data was not analyzed for this endpoint as there were no deaths.
Measure: Number; unit: Days
Arm/Group | Phase 3 Cohort 2 Pediatric (Placebo) | Phase 3 Cohort 2 Pediatric (1.2g IV) | Phase 3 Cohort 2 Pediatric (2.4g IV)
Number analyzed (Participants) | 1 | 121 | 70
Days | 0 | 0 | 0

71. Secondary Outcome: Proportion of Participants Requiring Mechanical Ventilation Due to COVID-19 (Ph3 Cohort 1- 1.2g vs Placebo)
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1 (Placebo) >= 18 | Phase 3 Cohort 1 (1.2g IV) >= 18
Number analyzed (Participants) | 748 | 736
Percentage of Participants | 0.3 [0.0 to 1.0] | 0.1 [0.0 to 0.8]

72. Secondary Outcome: Proportion of Participants Requiring Mechanical Ventilation Due to COVID-19 (Ph3 Cohort 1- 2.4g vs Placebo)
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Groups:
- Phase 3 Cohort 1 (Placebo): Phase 3 Cohort 1 Participants (Placebo)
Arm/Group | Phase 3 Cohort 1 (Placebo) | Phase 3 Cohort 1 (2.4g IV) >= 18
Number analyzed (Participants) | 1341 | 1355
Proportion of Participants | 0.4 [0.2 to 1.0] | 0.0007 [0.0 to 0.4]

73. Secondary Outcome: Proportion of Participants Requiring Mechanical Ventilation Due to COVID-19 (Phase 3 Cohort 2)
Description: Phase 3 (Cohort 2)
Time Frame: Through Day 29
Population: There were 0 events in this endpoint. Phase 3 Cohort 2 data was not analyzed for this endpoint as there were 0 events in in this cohort
Measure: Number; unit: Percent
Arm/Group | Phase 3 Cohort 2 Pediatric (Placebo) | Phase 3 Cohort 2 Pediatric (1.2g IV) | Phase 3 Cohort 2 Pediatric (2.4g IV)
Number analyzed (Participants) | 1 | 121 | 70
Percent | 0 | 0 | 0

74. Secondary Outcome: Change From Baseline in Viral Load at Each Visit, as Measured by RT-qPCR in Nasopharyngeal Swabs - (Phase 3 Cohort 1 - 1.2g vs. Placebo)
Description: Phase 3 Cohort 1
Time Frame: Baseline up to Day 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- Phase 3 Cohort 1 Placebo: Modified Full Analysis Set (mFAS) of Next Phase 3 Cohort 1 Participants
- Phase 3 Cohort 1 (1.2g IV): Phase 3 Cohort 1 Pediatric Participants Modified Full Analysis Set (mFAS)
Arm/Group | Phase 3 Cohort 1 Placebo | Phase 3 Cohort 1 (1.2g IV)
Number analyzed (Participants) | 748 | 736
log10 copies/mL
  Day 7: number analyzed (Participants) | 695 | 689
  Day 7 | -3.14 (1.964) | -3.90 (2.027)
  Day 15: number analyzed (Participants) | 672 | 686
  Day 15 | -5.01 (2.068) | -5.37 (2.098)
  Day 29: number analyzed (Participants) | 676 | 674
  Day 29 | -6.06 (1.976) | -6.32 (2.107)

75. Secondary Outcome: Change From Baseline in Viral Load at Each Visit, as Measured by RT-qPCR in Nasopharyngeal Swabs - (Phase 3 Cohort 1 - 2.4g vs. Placebo)
Description: Phase 3 Cohort 1
Time Frame: Baseline up to Day 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- Phase 3 Cohort 1 (2.4g IV): Phase 3 Cohort 1 Pediatric Participants Modified Full Analysis Set (mFAS)
Arm/Group | Phase 3 Cohort 1 Placebo | Phase 3 Cohort 1 (2.4g IV)
Number analyzed (Participants) | 1341 | 1355
log10 copies/mL
  Day 7: number analyzed (Participants) | 1227 | 1277
  Day 7 | -3.01 (1.951) | -3.89 (1.940)
  Day 15: number analyzed (Participants) | 1196 | 1259
  Day 15 | -5.02 (2.034) | -5.44 (2.104)
  Day 29: number analyzed (Participants) | 1207 | 1256
  Day 29 | -6.08 (1.943) | -6.19 (1.968)

76. Secondary Outcome: Change From Baseline in Viral Load at Each Visit, as Measured by RT-qPCR in Nasopharyngeal Swabs - (Phase 3 Cohort 2)
Description: Phase 3 Cohort 2
Time Frame: Baseline up to Day 29
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- Phase 3 Cohort 2 Placebo: Modified Full Analysis Set (mFAS) of Next Phase 3 Cohort 2 Participants
- Phase 3 Cohort 2 (1.2g IV): Phase 3 Cohort 2 (1.2g IV) Pediatric Participants Modified Full Analysis Set (mFAS)
- Phase 3 Cohort 2 (2.4g IV): Modified Full Analysis Set (mFAS) of Phase 3 Cohort (2.4g IV) Participants
Arm/Group | Phase 3 Cohort 2 Placebo | Phase 3 Cohort 2 (1.2g IV) | Phase 3 Cohort 2 (2.4g IV)
Number analyzed (Participants) | 1 | 121 | 70
log10 copies/mL
  Day 7: number analyzed (Participants) | 1 | 115 | 59
  Day 7 | -1.95 (NA) — Inadequate number of events to calculate standard deviation | -4.47 (2.522) | -5.23 (1.985)
  Day 15: number analyzed (Participants) | 1 | 115 | 58
  Day 15 | -4.50 (NA) — Inadequate number of events to calculate standard deviation | -6.10 (2.058) | -6.83 (1.940)
  Day 29: number analyzed (Participants) | 1 | 111 | 57
  Day 29 | -4.50 (NA) — Inadequate number of events to calculate standard deviation | -6.50 (1.930) | -7.06 (1.724)

77. Secondary Outcome: Time-weighted Average Change From Baseline in Viral Load (log10 Copies/mL), as Measured by Quantitative Reverse Transcription Quantitative Polymerase Chain Reaction (RT-qPCR) in Nasopharyngeal (NP) Swab Samples (Ph3 Cohort 1)
Description: Phase 3 (Cohort 1)
Time Frame: Baseline to Day 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- Phase 3 Cohort 1 Placebo: (Placebo) Participants who were ≥18 and not pregnant at time of randomization
- Phase 3 Cohort 1 2.4g IV: (2.4g IV) Participants who were ≥18 and not pregnant at time of randomization
- Phase 3 Cohort 1 8.0g IV: (8.0g IV) Participants who were ≥18 and not pregnant at time of randomization
Arm/Group | Phase 3 Cohort 1 Placebo | Phase 3 Cohort 1 2.4g IV | Phase 3 Cohort 1 8.0g IV
Number analyzed (Participants) | 571 | 603 | 608
log10 copies/mL | -1.46 (1.220) | -2.02 (1.021) | -2.05 (1.079)

78. Secondary Outcome: Time-weighted Average Change From Baseline in Viral Load (log10 Copies/mL), as Measured by Quantitative Reverse Transcription Quantitative Polymerase Chain Reaction (RT-qPCR) in Nasopharyngeal (NP) Swab Samples (Ph3 Cohort 2)
Description: Phase 3 (Cohort 2)
Time Frame: Baseline to Day 7
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- Phase 3 Cohort 2 Placebo: (Placebo) Participants who were less than 18 and not pregnant at time of randomization
- Phase 3 Cohort 2 (1.2g IV): (1.2g IV) Participants who were less than 18 and not pregnant at time of randomization
- Phase 3 Cohort 2 (2.4g IV): (2.4g IV) Participants who were less than 18 and not pregnant at time of randomization
Arm/Group | Phase 3 Cohort 2 Placebo | Phase 3 Cohort 2 (1.2g IV) | Phase 3 Cohort 2 (2.4g IV)
Number analyzed (Participants) | 1 | 117 | 62
log10 copies/mL | -0.97 (NA) — Unable to calculate SD due to number of participants analyzed | -2.49 (1.413) | -2.94 (1.435)

79. Secondary Outcome: Proportion of Participants With Viral Loads Below the Lower Limit of Detection at Each Visit - (Phase 2 Only)
Description: Next Phase 2 Symptomatic
Time Frame: Day 0, Day 5, Day 7, Day 15, Day 29
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Next Phase 2 (Placebo) | Next Phase 2 (2.4g IV) | Next Phase 2 (8.0g IV)
Number analyzed (Participants) | 150 | 142 | 145
Participants
  Day 0 (Baseline) | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 140 | 134 | 136
  Day 5 | 20 | 21 | 21
  Day 7: number analyzed (Participants) | 139 | 131 | 132
  Day 7 | 27 | 22 | 34
  Day 15: number analyzed (Participants) | 100 | 98 | 95
  Day 15 | 59 | 59 | 60
  Day 29: number analyzed (Participants) | 53 | 49 | 55
  Day 29 | 43 | 42 | 48

80. Secondary Outcome: Proportion of Participants With Viral Loads Below the Lower Limit of Quantitation at Each Visit - (Phase 2 Only)
Description: Next Phase 2 Symptomatic
Time Frame: Day 0, Day 5, Day 7, Day 15, Day 29
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Next Phase 2 (Placebo) | Next Phase 2 (2.4g IV) | Next Phase 2 (8.0g IV)
Number analyzed (Participants) | 150 | 142 | 145
Participants
  Day 0 (Baseline) | 6 | 5 | 6
  Day 5: number analyzed (Participants) | 140 | 134 | 136
  Day 5 | 25 | 26 | 28
  Day 7: number analyzed (Participants) | 139 | 131 | 132
  Day 7 | 38 | 38 | 47
  Day 15: number analyzed (Participants) | 100 | 98 | 95
  Day 15 | 68 | 72 | 74
  Day 29: number analyzed (Participants) | 53 | 49 | 55
  Day 29 | 50 | 46 | 51

81. Secondary Outcome: Number of Days of Hospitalization Due to COVID-19 (Ph3 Cohort 1) Placebo vs. 1.2g IV
Description: Phase 3 (Cohort 1)
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Phase 3 Cohort 1 (Placebo): Modified Full Analysis Set (mFAS) of Next Phase 3 Cohort 1 Participants
- Phase 3 Cohort 1 1.2g IV: Modified Full Analysis Set (mFAS) of Next Phase 3 Cohort 1 Participants 1.2g IV
Arm/Group | Phase 3 Cohort 1 (Placebo) | Phase 3 Cohort 1 1.2g IV
Number analyzed (Participants) | 62 | 736
Days | 10.0 (7.16) | 7.0 (8.04)

82. Secondary Outcome: Number of Days of Hospitalization Due to COVID-19 (Ph3 Cohort 1) Placebo vs. 2.4g IV
Description: Phase 3 (Cohort 1)
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Phase 3 Cohort 1 Pediatric (2.4g IV): Phase 3 Cohort 1 Pediatric (2.4g IV)
Arm/Group | Phase 3 Cohort 1 (Placebo) | Phase 3 Cohort 1 Pediatric (2.4g IV)
Number analyzed (Participants) | 24 | 736
Days | 8.4 (6.74) | 7.0 (8.04)

83. Secondary Outcome: Number of Days of Hospitalization Due to COVID-19 (Ph3 Cohort 2)
Description: Phase 3 (Cohort 2)
Time Frame: Through Day 29
Population: Participants <18 years old who, at baseline, were not pregnant, had symptomatic COVID-19, and had at least 1 risk factor for developing severe disease. No participants were hospitalized, therefore no hospitalizations days took place.
Groups:
- Phase 3 Cohort 2 Pediatric (Placebo): Phase 3 Cohort 2 Pediatric (Placebo) modified Full Analysis Set (mFAS)
- Phase 3 Cohort 2 Pediatric (1.2g IV): Phase 3 Cohort 2 Pediatric (1.2g IV) modified Full Analysis Set (mFAS)
- Phase 3 Cohort 2 Pediatric (2.4g IV): Phase 3 Cohort 2 Pediatric (2.4g IV) modified Full Analysis Set (mFAS)
Arm/Group | Phase 3 Cohort 2 Pediatric (Placebo) | Phase 3 Cohort 2 Pediatric (1.2g IV) | Phase 3 Cohort 2 Pediatric (2.4g IV)
Number analyzed (Participants) | 0 | 0 | 0

84. Secondary Outcome: Number of Days of Hospitalization Due to COVID-19 (Phase 2 Asymptomatic)
Description: Phase 2 Only
Time Frame: Up to Day 29
Population: Phase 2 asymptomatic cohort. No participants were hospitalized, therefore no hospitalizations days took place.
Arm/Group | Placebo | Phase 2 Asymptomatic: 2.4 IV | Phase 2 Asymptomatic: 8.0 IV
Number analyzed (Participants) | 0 | 0 | 0

85. Secondary Outcome: Proportion of Participants Admitted to an Intensive Care Unit (ICU) Due to COVID-19 - (Ph 3 Cohort 1) Placebo vs. 1.2g IV
Description: Phase 3 (Cohort 1)
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Groups:
- Phase 3 Cohort 1 (Placebo): Symptomatic Participants with COVID-19
- Phase 3 Cohort 1 (1.2g IV): Phase 3 Cohort 1 (1.2g IV)
Arm/Group | Phase 3 Cohort 1 (Placebo) | Phase 3 Cohort 1 (1.2g IV)
Number analyzed (Participants) | 748 | 736
Proportion of Participants | 0.9 [0.4 to 1.9] | 0.4 [0.1 to 1.2]

86. Secondary Outcome: Percentage of Participants Admitted to an Intensive Care Unit (ICU) Due to COVID-19 - (Ph 3 Cohort 1) Placebo vs. 2.4g IV
Description: Phase 3 (Cohort 1)
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Phase 3 Cohort 1 (2.4g IV): Phase 3 Cohort 1 (2.4g IV)
Arm/Group | Phase 3 Cohort 1 (Placebo) | Phase 3 Cohort 1 (2.4g IV)
Number analyzed (Participants) | 1341 | 1355
Percentage of Participants | 1.3 [0.8 to 2.1] | 0.4 [0.2 to 1.0]

87. Secondary Outcome: Proportion of Participants Admitted to an Intensive Care Unit (ICU) Due to COVID-19 - (Ph 3 Cohort 2)
Description: Phase 3 (Cohort 2)
Time Frame: Through Day 29
Population: as for outcome 29
Measure: Number; unit: Participants
Arm/Group | Phase 3 Cohort 2 Pediatric (Placebo) | Phase 3 Cohort 2 Pediatric (1.2g IV) | Phase 3 Cohort 2 Pediatric (2.4g IV)
Number analyzed (Participants) | 1 | 121 | 70
Participants | 0 | 0 | 0

88. Secondary Outcome: Proportion of Participants Admitted to an Intensive Care Unit (ICU) Due to COVID-19 - (Next Phase 2) #87
Description: Next Phase 2
Time Frame: Through Day 29
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Next Phase 2 (Placebo) | Next Phase 2 (2.4g IV) | Next Phase 2 (8.0g IV)
Number analyzed (Participants) | 150 | 142 | 145
Participants | 0 | 0 | 0

89. Secondary Outcome: Total Number of COVID-19-related Medically-attended Visits (Phase 3 Cohort 1) Placebo vs. 1.2g
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Number of Visits
Groups:
- Placebo: Placebo mFAS (modified Full Analysis Set)
- Phase 3 Cohort 1 1.2g IV: Phase 3 Cohort 1 1.2 g IV mFAS (modified Full Analysis Set)
Arm/Group | Placebo | Phase 3 Cohort 1 1.2g IV
Number analyzed (Participants) | 51 | 20
Number of Visits | 1.1 (0.27) | 1.2 (0.52)

90. Secondary Outcome: Total Number of COVID-19-related Medically-attended Visits (Phase 3 Cohort 1) Placebo vs. 2.4g
Description: Phase 3 Cohort 1
Time Frame: Through Day 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Number of Visits
Groups:
- Phase 3 Cohort 1 2.4g IV: Phase 3 Cohort 1 2.4g IV mFAS (modified Full Analysis Set)
Arm/Group | Placebo | Phase 3 Cohort 1 2.4g IV
Number analyzed (Participants) | 109 | 43
Number of Visits | 1.2 (0.41) | 1.0 (0.15)

91. Secondary Outcome: Total Number of COVID-19-related Medically-attended Visits (Phase 3 Cohort 2)
Description: Phase 3 Cohort 2
Time Frame: Through Day 29
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Number of Visits
Groups:
- Phase 3 Cohort 2 1.2g IV: Phase 3 Cohort 2 1.2g IV mFAS (modified Full Analysis Set)
- Phase 3 Cohort 2 2.4g IV: Phase 3 Cohort 2 2.4g IV mFAS (modified Full Analysis Set)
Arm/Group | Placebo | Phase 3 Cohort 2 1.2g IV | Phase 3 Cohort 2 2.4g IV
Number analyzed (Participants) | 1 | 121 | 70
Number of Visits | 1.0 (0.0) | 1.0 (NA) — too small a number of data points to calculate | 1.0 (0.0)

ADVERSE EVENTS:
Time Frame: From first dose to end of study (approx. 8 months)
Groups:
- Phase 1 Symptomatic Placebo; Phase 2 Symptomatic Placebo: Placebo of R10933 + R10987 Adult Symptomatic Participants with COVID-19
- Phase 1 Symptomatic R10933+R10987 2.4g IV; Phase 2 Symptomatic R10933+R10987 2.4g IV: 2.4g of R10933 + R10987 Adult Symptomatic Participants with COVID-19
- Phase 1 Symptomatic R10933+R10987 8.0g IV; Phase 2 Symptomatic R10933+R10987 8.0g IV: 8.0g of R10933 + R10987 Adult Symptomatic Participants with COVID-19
- Phase 3 Age>=18 Placebo: Placebo of R10933 + R10987 Participants >=18 with COVID-19, not pregnant at randomization
- Phase 3 Age>=18 R10933+R10987 1.2g IV: 1.2g of R10933 + R10987 Participants >=18 with COVID-19, not pregnant at randomization
- Phase 3 Age>=18 R10933+R10987 2.4g IV: 2.4g of R10933 + R10987 Participants >=18 with COVID-19, not pregnant at randomization
- Phase 3 Age>=18 R10933+R10987 8.0g IV: 8.0g of R10933 + R10987 Participants >=18 with COVID-19, not pregnant at randomization
- Phase 3 Age<18 Placebo: Placebo of R10933 + R10987 Participants <18 with COVID-19, not pregnant at randomization
- Phase 3 Age<18 R10933+R10987 1.2g IV: 1.2g of R10933 + R10987 Participants <18 with COVID-19
- Phase 3 Age<18 R10933+R10987 2.4g IV: 2.4g of R10933 + R10987 Participants <18 with COVID-19
- Phase 3 Pregnant R10933+R10987 1.2g IV: 1.2g of R10933 + R10987 Participants who are pregnant with COVID-19
- Phase 3 Pregnant R10933+R10987 2.4g IV: 2.4g of R10933 + R10987 Participants who are pregnant with COVID-19
Arm/Group | Phase 1 Symptomatic Placebo | Phase 1 Symptomatic R10933+R10987 2.4g IV | Phase 1 Symptomatic R10933+R10987 8.0g IV | Phase 2 Symptomatic Placebo | Phase 2 Symptomatic R10933+R10987 2.4g IV | Phase 2 Symptomatic R10933+R10987 8.0g IV | Phase 2 Asymptomatic Placebo | Phase 2 Asymptomatic R10933+R10987 2.4g IV | Phase 2 Asymptomatic R10933+R10987 8.0g IV | Phase 3 Age>=18 Placebo | Phase 3 Age>=18 R10933+R10987 1.2g IV | Phase 3 Age>=18 R10933+R10987 2.4g IV | Phase 3 Age>=18 R10933+R10987 8.0g IV | Phase 3 Age<18 Placebo | Phase 3 Age<18 R10933+R10987 1.2g IV | Phase 3 Age<18 R10933+R10987 2.4g IV | Phase 3 Pregnant Placebo | Phase 3 Pregnant R10933+R10987 1.2g IV | Phase 3 Pregnant R10933+R10987 2.4g IV
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22 | 0/23 | 0/238 | 0/236 | 0/237 | 0/73 | 0/74 | 0/75 | 11/2347 | 2/2130 | 4/3157 | 0/1012 | 0/2 | 0/129 | 0/71 | 0/2 | 0/43 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/22 | 0/23 | 6/238 | 3/236 | 2/237 | 0/73 | 0/74 | 0/75 | 103/2347 | 39/2130 | 52/3157 | 19/1012 | 0/2 | 3/129 | 0/71 | 0/2 | 11/43 | 7/35
Other Adverse Events (participants affected / at risk) | 0/24 | 0/22 | 0/23 | 2/238 | 1/236 | 1/237 | 0/73 | 0/74 | 0/75 | 16/2347 | 16/2130 | 19/3157 | 4/1012 | 1/2 | 0/129 | 1/71 | 0/2 | 5/43 | 3/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Symptomatic Placebo (N=24) | Phase 1 Symptomatic R10933+R10987 2.4g IV (N=22) | Phase 1 Symptomatic R10933+R10987 8.0g IV (N=23) | Phase 2 Symptomatic Placebo (N=238) | Phase 2 Symptomatic R10933+R10987 2.4g IV (N=236) | Phase 2 Symptomatic R10933+R10987 8.0g IV (N=237) | Phase 2 Asymptomatic Placebo (N=73) | Phase 2 Asymptomatic R10933+R10987 2.4g IV (N=74) | Phase 2 Asymptomatic R10933+R10987 8.0g IV (N=75) | Phase 3 Age>=18 Placebo (N=2347) | Phase 3 Age>=18 R10933+R10987 1.2g IV (N=2130) | Phase 3 Age>=18 R10933+R10987 2.4g IV (N=3157) | Phase 3 Age>=18 R10933+R10987 8.0g IV (N=1012) | Phase 3 Age<18 Placebo (N=2) | Phase 3 Age<18 R10933+R10987 1.2g IV (N=129) | Phase 3 Age<18 R10933+R10987 2.4g IV (N=71) | Phase 3 Pregnant Placebo (N=2) | Phase 3 Pregnant R10933+R10987 1.2g IV (N=43) | Phase 3 Pregnant R10933+R10987 2.4g IV (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia neonatal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve calcification (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal atresia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniosynostosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macrocephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever neonatal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 20 (21) | 3 (3) | 9 (9) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 19 (21) | 5 (5) | 6 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 19 (20) | 5 (5) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Continuous glucose monitoring (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyporesponsive to stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perinatal depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
May-Thurner syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Symptomatic Placebo (N=24) | Phase 1 Symptomatic R10933+R10987 2.4g IV (N=22) | Phase 1 Symptomatic R10933+R10987 8.0g IV (N=23) | Phase 2 Symptomatic Placebo (N=238) | Phase 2 Symptomatic R10933+R10987 2.4g IV (N=236) | Phase 2 Symptomatic R10933+R10987 8.0g IV (N=237) | Phase 2 Asymptomatic Placebo (N=73) | Phase 2 Asymptomatic R10933+R10987 2.4g IV (N=74) | Phase 2 Asymptomatic R10933+R10987 8.0g IV (N=75) | Phase 3 Age>=18 Placebo (N=2347) | Phase 3 Age>=18 R10933+R10987 1.2g IV (N=2130) | Phase 3 Age>=18 R10933+R10987 2.4g IV (N=3157) | Phase 3 Age>=18 R10933+R10987 8.0g IV (N=1012) | Phase 3 Age<18 Placebo (N=2) | Phase 3 Age<18 R10933+R10987 1.2g IV (N=129) | Phase 3 Age<18 R10933+R10987 2.4g IV (N=71) | Phase 3 Pregnant Placebo (N=2) | Phase 3 Pregnant R10933+R10987 1.2g IV (N=43) | Phase 3 Pregnant R10933+R10987 2.4g IV (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 16 (16) | 16 (17) | 12 (12) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Nasal and saliva sample collection was discontinued early in the study because nasopharyngeal samples were determined to be more reliable for quantitative analysis, as such endpoints related to nasal or saliva samples were not analyzed. The Phase 1/2 SAP does not specify any analyses related to nasal and saliva samples collections

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (3):
  • Study Protocol (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT04425629/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT04425629/SAP_002.pdf
  • Informed Consent Form (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT04425629/ICF_000.pdf